CLINICAL TRIAL: NCT00372112
Title: A 2-wk Study to Evaluate the Safety, Tolerability,Pharmacodynamics and Pharmacokinetics of GW642444H(100 Administered Once Daily in the Morning Via DISKUS™ Dry-powder Inhaler)Compared With SEREVENT(Salmeterol)(50mcg Administered Twice Daily Via DISKUS Dry-powder Inhaler)and Placebo in Subject w/COPD
Brief Title: A Study To Assess The Safety And Tolerability Of GW642444 In Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2C108562
Record Dates: First submitted 2006-09-04; First posted 2006-09-06 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease (COPD); COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 100 mcg GW642444H (Active Comparator): Twice daily in the morning.
  Interventions: Drug: GW642444
- 400 mcg GW642444H (Active Comparator): Twice daily in the morning.
  Interventions: Drug: GW642444
- 50 mcg salmeterol (Active Comparator): Twice daily.
  Interventions: Drug: GW642444
- placebo (Placebo Comparator): Twice daily
  Interventions: Drug: GW642444; Other: Placebo

INTERVENTIONS:
Drug: GW642444 — GW642444H
Other: Placebo — Placebo administered twice daily
  Arms: placebo

SUMMARY:
The compound GW642444 has previously been found to be well tolerated with no significant side effects in subjects with asthma and healthy volunteers. This study will assess the safety and tolerability of GW642444 in subjects with COPD in order to obtain information to support dosing in a broader population of subjects with COPD

DETAILED DESCRIPTION:
A multicentre, randomised, placebo-controlled, double-blind, 4-arm parallel-group, 2-week study to evaluate the safety, tolerability, pharmacodynamics and pharmacokinetics of GW642444H (100 administered once daily in the morning via DISKUS™ dry-powder inhaler) compared with SEREVENT (salmeterol) (50mcg administered twice daily via DISKUS dry-powder inhaler) and placebo in subjects with moderate COPD.

ELIGIBILITY:
Inclusion criteria:

* females must be of non-childbearing potential
* moderately severe COPD

Exclusion criteria:

* Subjects with a main diagnosis of asthma
* subjects with poorly controlled COPD
* subjects with significant heart, renal, endocrine, psychiatric, immunological or neurological disease.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2006-11-03 (Actual); Primary Completion 2007-05-01 (Actual); Study Completion 2007-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- Australia (2):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Nedlands, Western Australia
- Bulgaria (2):
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
- Germany (3):
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
- Netherlands (2):
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Hoorn
- New Zealand (2):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Tauranga
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: B2C108562 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: B2C108562 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: B2C108562 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: B2C108562 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: B2C108562 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: B2C108562 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: B2C108562 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned on 80 male or female participants with moderate chronic obstructive pulmonary disease (COPD), aged 40 years or older from 03 November 2006 to 10 May 2007, across 14 centers of 6 countries (10 centers in Europe, 2 centers in Australia and 2 centers in New Zealand).
Pre-assignment Details: Out of 145 participants screened, 77 were screen failures and remaining 68 participants were randomized in the study to receive placebo, GW642444H (100 microgram [mcg] or 400 mcg once daily or Salmeterol 50 mcg twice daily (BD) via the DISKUS® dry powder inhaler (DPI).
Groups:
- Placebo: Participants received oral inhalations of matching placebo via DISKUS DPI, BD for 2 weeks of treatment period. Participants were provided with 3 inhalers (Inhaler A, B and C) to maintain the blinding. Participants received morning dose of 1 inhalation of placebo from Inhaler A and 3 inhalations of placebo from Inhaler B and evening dose of 1 inhalation of placebo from Inhaler C. Inhaled short acting beta-agonists, ipratropium bromide was provided as rescue medication throughout the study.
- GW642444 100 mcg Once Daily: Participants received oral inhalations of GW642444 100 mcg via DISKUS DPI, once daily for 2 weeks of treatment period. Participants were provided with 3 inhalers (Inhaler A, B and C) to maintain the blinding. Participants received morning dose of 1 inhalation of GW642444 100 mcg from Inhaler A and 3 inhalations of placebo from Inhaler B and evening dose of 1 inhalation of placebo from Inhaler C. Inhaled short acting beta-agonists, ipratropium bromide was provided as rescue medication throughout the study.
- GW642444 400 mcg Once Daily: Participants received oral inhalations of GW642444 100 mcg via DISKUS DPI, once daily for 2 weeks of treatment period. Participants were provided with 3 inhalers (Inhaler A, B and C) to maintain the blinding. Participants received morning dose of 1 inhalation of GW642444 100 mcg from Inhaler A and 3 inhalations of GW642444 100 mcg (3 inhalations x GW642444 100 mcg) from Inhaler B and evening dose of 1 inhalation of placebo from Inhaler C. Inhaled short acting beta-agonists, ipratropium bromide was provided as rescue medication throughout the study.
- Salmeterol 50 mcg BD: Participants received oral inhalations of salmeterol 50 mcg via DISKUS DPI, BD for 2 weeks of treatment period. Participants were provided with 3 inhalers (Inhaler A, B and C) to maintain the blinding. Participants received morning dose of 1 inhalation of salmeterol 50 mcg from Inhaler A and 3 inhalations of placebo from Inhaler B and evening dose of 1 inhalation of salmeterol 50 mcg from Inhaler C. Inhaled short acting beta-agonists, ipratropium bromide was provided as rescue medication throughout the study.
Period: Overall Study
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Started | 17 | 16 | 17 | 18
Completed | 16 | 15 | 13 | 14
Not Completed | 1 | 1 | 4 | 4
Not completed — Adverse Event | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Exacerbation | 0 | 0 | 0 | 1
Not completed — PR >240 at Visit 3 | 0 | 0 | 0 | 1
Not completed — Hepatitis B | 1 | 0 | 0 | 0
Not completed — Other-protocol violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD | Total
Number analyzed (Participants) | 17 | 16 | 17 | 18 | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (8.79) | 65.8 (9.06) | 66.6 (9.16) | 60.2 (7.37) | 63.4 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 5 | 9 | 24
  Male | 13 | 10 | 12 | 9 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 2
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 16 | 15 | 17 | 18 | 66
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Time Frame: Up to Follow-up (17 days)
Population: Safety Population comprised of all participants who were randomized and received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
Participants
  Any AE | 4 | 5 | 7 | 6
  Any SAE | 0 | 0 | 1 | 1

2. Secondary Outcome: Change From Baseline in Pre-dose Weighted Mean Heart Rate (HR) Derived From 28.5 Hour (h) Ambulatory Blood Pressure Monitoring (ABPM) at Day 7 and 14
Description: HR was measured using 28.5h ABPM on Day 1, Day 7 and Day 14. Baseline was defined as the pre-dose weighted mean of Day 1. Weighted mean was calculated by calculating the area under curve (AUC) of measurements made pre-dose on each day, and then dividing by the relevant time interval. AUC was calculated using the trapezoidal rule. The weighted mean change from Baseline was the average AUC minus Baseline (AAUCMB).
Time Frame: Baseline (Day 1, pre-dose) up to Day 14
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
Beats per minute (bpm)
  Day 7: number analyzed (Participants) | 12 | 14 | 11 | 11
  Day 7 | 4.60 (5.689) | 0.18 (7.253) | 0.17 (6.443) | 0.95 (8.793)
  Day 14: number analyzed (Participants) | 12 | 13 | 10 | 9
  Day 14 | 1.13 (7.151) | -1.31 (9.724) | 4.29 (9.646) | -0.22 (7.345)

3. Secondary Outcome: Change From Baseline in 0-4 h Weighted Mean HR Derived From 28.5 h ABPM at Day 1, 2, 7, 8, 14 and 15
Description: HR was measured using 28.5 h ABPM on Day 1 (continued till Day 2), Day 7 (continued till Day 8) and Day 14 (continued till Day 15). Baseline was defined as the pre-dose weighted mean of Day 1. Weighted mean was calculated by calculating the AUC of measurements made 0-4 h post-dose on Day 1, 2, 7, 8, 14 and 15 and then dividing by the relevant time interval. AUC was calculated using the trapezoidal rule. The weighted mean change from Baseline was the AAUCMB.
Time Frame: Baseline (Day 1, pre-dose) up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
bpm
  Day 1: number analyzed (Participants) | 13 | 16 | 15 | 14
  Day 1 | 2.14 (2.134) | 4.25 (1.848) | 7.47 (1.993) | 4.63 (2.020)
  Day 2: number analyzed (Participants) | 12 | 16 | 15 | 12
  Day 2 | 1.01 (2.208) | 0.63 (1.838) | 5.37 (1.987) | 5.61 (2.138)
  Day 7: number analyzed (Participants) | 12 | 14 | 11 | 11
  Day 7 | 8.21 (2.357) | 3.95 (2.051) | 7.76 (2.403) | 6.75 (2.324)
  Day 8: number analyzed (Participants) | 12 | 14 | 12 | 11
  Day 8 | 1.11 (2.341) | 1.27 (2.046) | 9.41 (2.377) | 4.94 (2.317)
  Day 14: number analyzed (Participants) | 12 | 13 | 10 | 9
  Day 14 | 3.64 (2.307) | 2.54 (2.037) | 10.42 (2.528) | 6.92 (2.476)
  Day 15: number analyzed (Participants) | 12 | 14 | 10 | 11
  Day 15 | 2.17 (2.460) | 1.04 (2.138) | 5.76 (2.666) | 4.28 (2.440)
Statistical Analysis 1: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for 0-4 h at Day 1; Test type: Superiority; Mean Difference (Net) = 2.11, 95% CI 2-sided [-3.48 to 7.70]
Statistical Analysis 2: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for 0-4 h at Day 1; Test type: Superiority; Mean Difference (Net) = 5.33, 95% CI 2-sided [-0.41 to 11.07]
Statistical Analysis 3: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for 0-4 h at Day 1; Test type: Superiority; Mean Difference (Net) = 2.49, 95% CI 2-sided [-3.35 to 8.33]
Statistical Analysis 4: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for 0-4 h at Day 2; Test type: Superiority; Mean Difference (Net) = -0.38, 95% CI 2-sided [-6.11 to 5.36]
Statistical Analysis 5: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for 0-4 h at Day 2; Test type: Superiority; Mean Difference (Net) = 4.36, 95% CI 2-sided [-1.57 to 10.29]
Statistical Analysis 6: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for 0-4 h at Day 2; Test type: Superiority; Mean Difference (Net) = 4.60, 95% CI 2-sided [-1.45 to 10.65]
Statistical Analysis 7: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for 0-4 h at Day 7; Test type: Superiority; Mean Difference (Net) = -4.25, 95% CI 2-sided [-10.44 to 1.93]
Statistical Analysis 8: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for 0-4 h at Day 7; Test type: Superiority; Mean Difference (Net) = -0.45, 95% CI 2-sided [-7.22 to 6.32]
Statistical Analysis 9: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for 0-4 h at Day 7; Test type: Superiority; Mean Difference (Net) = -1.46, 95% CI 2-sided [-8.25 to 5.33]
Statistical Analysis 10: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for 0-4 h at Day 8; Test type: Superiority; Mean Difference (Net) = 0.16, 95% CI 2-sided [-5.98 to 6.29]
Statistical Analysis 11: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for 0-4 h at Day 8; Test type: Superiority; Mean Difference (Net) = 8.30, 95% CI 2-sided [1.52 to 15.08]
Statistical Analysis 12: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for 0-4 h at Day 8; Test type: Superiority; Mean Difference (Net) = 3.82, 95% CI 2-sided [-2.85 to 10.50]
Statistical Analysis 13: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for 0-4 h at Day 14; Test type: Superiority; Mean Difference (Net) = -1.09, 95% CI 2-sided [-7.16 to 4.97]
Statistical Analysis 14: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for 0-4 h at Day 14; Test type: Superiority; Mean Difference (Net) = 6.78, 95% CI 2-sided [-0.11 to 13.66]
Statistical Analysis 15: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for 0-4 h at Day 14; Test type: Superiority; Mean Difference (Net) = 3.29, 95% CI 2-sided [-3.58 to 10.15]
Statistical Analysis 16: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for 0-4 h at Day 15; Test type: Superiority; Mean Difference (Net) = -1.12, 95% CI 2-sided [-7.64 to 5.40]
Statistical Analysis 17: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for 0-4 h at Day 15; Test type: Superiority; Mean Difference (Net) = 3.59, 95% CI 2-sided [-3.71 to 10.89]
Statistical Analysis 18: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for 0-4 h at Day 15; Test type: Superiority; Mean Difference (Net) = 2.11, 95% CI 2-sided [-4.96 to 9.18]

4. Secondary Outcome: Change From Baseline in 0-24 h Weighted Mean HR Derived From 28.5 ABPM at Day 7 and 14
Description: HR was measured using 28.5 h ABPM on Day 1, Day 7 and Day 14. Baseline was defined as the pre-dose weighted mean of Day 1. Weighted mean was calculated by calculating the AUC of measurements made 0-24 h post-dose on Day 7 and 14, and then dividing by the relevant time interval. AUC was calculated using the trapezoidal rule. The weighted mean change from Baseline was the AAUCMB.
Time Frame: Baseline (Day 1, pre-dose) up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
bpm
  Day 7: number analyzed (Participants) | 12 | 14 | 11 | 11
  Day 7 | 6.50 (6.696) | 3.07 (7.261) | 7.16 (6.567) | 6.47 (6.885)
  Day 14: number analyzed (Participants) | 12 | 13 | 10 | 9
  Day 14 | 2.77 (7.495) | 1.84 (7.389) | 9.23 (8.173) | 5.87 (6.420)

5. Secondary Outcome: Change From Baseline in Maximum HR During 0-4 h Derived From 28.5 h ABPM at Day 1, 2, 7, 8, 14 and 15
Description: HR was measured using 28.5 h ABPM on Day 1 (continued till Day 2), Day 7 (continued till Day 8) and Day 14 (continued till Day 15). For the calculation of 0-4 h maximum change from Baseline, measurements post-dose up to 6 h (actual time) was included. Baseline was defined as the pre-dose weighted mean of Day 1. Maximum change from Baseline was calculated by subtracting the Baseline value (weighted mean pre-dose Day 1) from the maximum assessment value (during 0-4 h) of the individual post-Baseline time points.
Time Frame: Baseline (Day 1, pre-dose) up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
bpm
  Day 1: number analyzed (Participants) | 14 | 16 | 15 | 15
  Day 1 | 20.6 (3.71) | 22.7 (3.35) | 23.5 (3.61) | 20.5 (3.51)
  Day 2: number analyzed (Participants) | 12 | 16 | 15 | 14
  Day 2 | 9.7 (3.17) | 11.9 (2.66) | 15.5 (2.88) | 11.3 (2.90)
  Day 7: number analyzed (Participants) | 13 | 15 | 12 | 11
  Day 7 | 26.8 (4.21) | 21.9 (3.68) | 25.0 (4.37) | 22.0 (4.36)
  Day 8: number analyzed (Participants) | 13 | 15 | 12 | 11
  Day 8 | 9.0 (2.85) | 12.4 (2.49) | 19.8 (2.96) | 12.1 (2.95)
  Day 14: number analyzed (Participants) | 13 | 15 | 10 | 11
  Day 14 | 26.1 (3.73) | 19.0 (3.25) | 31.5 (4.29) | 23.2 (3.86)
  Day 15: number analyzed (Participants) | 13 | 15 | 11 | 11
  Day 15 | 10.2 (3.04) | 10.5 (2.65) | 17.0 (3.27) | 14.6 (3.13)
Statistical Analysis 1: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for 0-4 h maximum HR at Day 1; Test type: Superiority; Mean Difference (Net) = 2.1, 95% CI 2-sided [-7.7 to 12.0]
Statistical Analysis 2: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for 0-4 h maximum HR at Day 1; Test type: Superiority; Mean Difference (Net) = 3.0, 95% CI 2-sided [-7.2 to 13.1]
Statistical Analysis 3: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for 0-4 h maximum HR at Day 1; Test type: Superiority; Mean Difference (Net) = 0.0, 95% CI 2-sided [-10.2 to 10.1]
Statistical Analysis 4: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for 0-4 h maximum HR at Day 2; Test type: Superiority; Mean Difference (Net) = 2.2, 95% CI 2-sided [-6.1 to 10.4]
Statistical Analysis 5: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for 0-4 h maximum HR at Day 2; Test type: Superiority; Mean Difference (Net) = 5.8, 95% CI 2-sided [-2.8 to 14.3]
Statistical Analysis 6: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for 0-4 h maximum HR at Day 2; Test type: Superiority; Mean Difference (Net) = 1.6, 95% CI 2-sided [-6.9 to 10.1]
Statistical Analysis 7: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for 0-4 h maximum HR at Day 7; Test type: Superiority; Mean Difference (Net) = -4.9, 95% CI 2-sided [-16.1 to 6.2]
Statistical Analysis 8: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for 0-4 h maximum HR at Day 7; Test type: Superiority; Mean Difference (Net) = -1.9, 95% CI 2-sided [-14.0 to 10.2]
Statistical Analysis 9: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for 0-4 h maximum HR at Day 7; Test type: Superiority; Mean Difference (Net) = -4.8, 95% CI 2-sided [-17.1 to 7.5]
Statistical Analysis 10: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for 0-4 h maximum HR at Day 8; Test type: Superiority; Mean Difference (Net) = 3.4, 95% CI 2-sided [-4.1 to 10.9]
Statistical Analysis 11: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for 0-4 h maximum HR at Day 8; Test type: Superiority; Mean Difference (Net) = 10.8, 95% CI 2-sided [2.6 to 19.0]
Statistical Analysis 12: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for 0-4 h maximum HR at Day 8; Test type: Superiority; Mean Difference (Net) = 3.1, 95% CI 2-sided [-5.2 to 11.4]
Statistical Analysis 13: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for 0-4 h maximum HR at Day 14; Test type: Superiority; Mean Difference (Net) = -7.2, 95% CI 2-sided [-17.0 to 2.7]
Statistical Analysis 14: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for 0-4 h maximum HR at Day 14; Test type: Superiority; Mean Difference (Net) = 5.4, 95% CI 2-sided [-6.0 to 16.8]
Statistical Analysis 15: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for 0-4 h maximum HR at Day 14; Test type: Superiority; Mean Difference (Net) = -2.9, 95% CI 2-sided [-13.8 to 8.0]
Statistical Analysis 16: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for 0-4 h maximum HR at Day 15; Test type: Superiority; Mean Difference (Net) = 0.2, 95% CI 2-sided [-7.8 to 8.3]
Statistical Analysis 17: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for 0-4 h maximum HR at Day 15; Test type: Superiority; Mean Difference (Net) = 6.8, 95% CI 2-sided [-2.1 to 15.6]
Statistical Analysis 18: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for 0-4 h maximum HR at Day 15; Test type: Superiority; Mean Difference (Net) = 4.4, 95% CI 2-sided [-4.5 to 13.3]

6. Secondary Outcome: Mean Weighted Mean HR at 0-4 h, Weighted Mean HR at 0-24 h and Maximum HR at 0-4 h Derived From 28.5 h ABPM
Description: HR was measured using 28.5 h ABPM. Weighted mean HR at 0-4 h was obtained from measurements made over 0-4 h post-dose on Day 1, 2, 7, 8, 14 and 15. Weighted mean HR at 0-24 h was obtained from measurements made 0-24 h post-dose on Day 1, 7 and 14. Maximum HR at 0-4 h was obtained from measurements made over 0-4 h post-dose on Day 1, 2, 7, 8, 14 and 15. Baseline was defined as the pre-dose weighted mean of Day 1.
Time Frame: Day 1 up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
bpm
  Weighted mean HR 0-4, Day 1: number analyzed (Participants) | 13 | 16 | 15 | 14
  Weighted mean HR 0-4, Day 1 | 70.08 (10.722) | 72.23 (12.766) | 73.03 (13.251) | 77.50 (10.092)
  Weighted mean HR 0-4, Day 2: number analyzed (Participants) | 13 | 16 | 17 | 15
  Weighted mean HR 0-4, Day 2 | 71.07 (14.743) | 68.24 (10.081) | 70.47 (11.771) | 77.12 (11.461)
  Weighted mean HR 0-4, Day 7: number analyzed (Participants) | 14 | 14 | 13 | 13
  Weighted mean HR 0-4, Day 7 | 78.69 (12.493) | 73.01 (12.943) | 73.63 (10.354) | 78.44 (13.191)
  Weighted mean HR 0-4, Day 8: number analyzed (Participants) | 14 | 14 | 14 | 14
  Weighted mean HR 0-4, Day 8 | 73.82 (15.927) | 70.17 (11.353) | 73.20 (13.379) | 77.76 (13.003)
  Weighted mean HR 0-4, Day 14: number analyzed (Participants) | 15 | 13 | 11 | 12
  Weighted mean HR 0-4, Day 14 | 76.49 (12.635) | 71.14 (11.771) | 73.74 (11.469) | 80.39 (10.801)
  Weighted mean HR 0-4, Day 15: number analyzed (Participants) | 15 | 14 | 12 | 14
  Weighted mean HR 0-4, Day 15 | 75.64 (18.666) | 68.82 (12.980) | 73.00 (11.033) | 77.60 (10.298)
  Weighted mean HR 0-24, Day 1: number analyzed (Participants) | 13 | 16 | 15 | 14
  Weighted mean HR 0-24, Day 1 | 70.07 (10.079) | 72.33 (11.592) | 71.83 (11.772) | 78.53 (8.525)
  Weighted mean HR 0-24, Day 7: number analyzed (Participants) | 14 | 14 | 13 | 13
  Weighted mean HR 0-24, Day 7 | 75.83 (11.085) | 72.35 (11.046) | 74.05 (11.298) | 78.18 (9.649)
  Weighted mean HR 0-24, Day 14: number analyzed (Participants) | 15 | 13 | 11 | 12
  Weighted mean HR 0-24, Day 14 | 75.72 (11.473) | 70.45 (10.977) | 72.42 (10.097) | 78.93 (8.054)
  Maximum HR 0-4 h, Day 1: number analyzed (Participants) | 16 | 16 | 17 | 18
  Maximum HR 0-4 h, Day 1 | 94.9 (18.38) | 90.3 (17.72) | 88.6 (13.91) | 92.7 (13.90)
  Maximum HR 0-4 h, Day 2: number analyzed (Participants) | 14 | 16 | 17 | 17
  Maximum HR 0-4 h, Day 2 | 82.4 (17.80) | 79.4 (15.90) | 79.5 (16.07) | 86.3 (14.03)
  Maximum HR 0-4 h, Day 7: number analyzed (Participants) | 16 | 15 | 14 | 14
  Maximum HR 0-4 h, Day 7 | 97.9 (13.76) | 90.5 (18.85) | 88.7 (17.07) | 94.6 (14.86)
  Maximum HR 0-4 h, Day 8: number analyzed (Participants) | 15 | 15 | 14 | 14
  Maximum HR 0-4 h, Day 8 | 82.2 (19.23) | 80.6 (18.06) | 82.0 (16.14) | 86.9 (14.31)
  Maximum HR 0-4 h, Day 14: number analyzed (Participants) | 16 | 15 | 12 | 14
  Maximum HR 0-4 h, Day 14 | 95.2 (12.16) | 87.0 (14.68) | 92.9 (20.08) | 96.2 (12.21)
  Maximum HR 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 13 | 14
  Maximum HR 0-4 h, Day 15 | 84.8 (19.24) | 78.7 (16.37) | 82.6 (10.95) | 88.7 (13.90)

7. Secondary Outcome: Mean Hourly HR 0-24 h at Day 1, 7 and 14
Description: HR was measured using 28.5 h ABPM. The assessments were analyzed hourly as 0-1 h, 1-2 h, 2-3 h, 3-4 h, 4-5 h, 5-6 h, 6-7 h, 7-8 h, 8-9 h, 9-10 h, 10-11 h, 11-12 h, 12-13 h, 13-14 h, 14-15 h, 15-16 h, 16-17 h, 17-18 h, 18-19 h, 19-20 h, 20-21 h, 21-22 h, 22-23 h and 23-24 h at Day 1, Day 7 and Day 14.
Time Frame: Day 1 up to Day 14
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
bpm
  Day 1, 0-1 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 0-1 h | 68.20 (12.487) | 68.38 (11.616) | 72.51 (14.025) | 73.48 (10.304)
  Day 1, 1-2 h: number analyzed (Participants) | 15 | 16 | 15 | 17
  Day 1, 1-2 h | 68.84 (14.022) | 69.89 (13.158) | 73.50 (14.366) | 72.88 (10.279)
  Day 1, 2-3 h: number analyzed (Participants) | 15 | 12 | 16 | 14
  Day 1, 2-3 h | 72.87 (18.200) | 66.83 (14.839) | 70.09 (16.775) | 76.29 (11.530)
  Day 1, 3-4 h: number analyzed (Participants) | 13 | 15 | 15 | 16
  Day 1, 3-4 h | 68.69 (14.133) | 72.29 (15.321) | 70.43 (12.784) | 75.09 (10.270)
  Day 1, 4-5 h: number analyzed (Participants) | 14 | 16 | 16 | 16
  Day 1, 4-5 h | 80.07 (22.088) | 74.82 (17.671) | 77.72 (13.937) | 83.50 (12.022)
  Day 1, 5-6 h: number analyzed (Participants) | 14 | 14 | 15 | 15
  Day 1, 5-6 h | 90.46 (17.075) | 79.68 (16.218) | 83.83 (11.544) | 84.77 (16.272)
  Day 1, 6-7 h: number analyzed (Participants) | 14 | 15 | 16 | 14
  Day 1, 6-7 h | 85.64 (16.974) | 78.23 (17.370) | 76.54 (12.801) | 81.46 (11.896)
  Day 1, 7-8 h: number analyzed (Participants) | 12 | 16 | 15 | 15
  Day 1, 7-8 h | 81.67 (16.306) | 78.28 (15.727) | 78.14 (15.623) | 81.40 (11.960)
  Day 1, 8-9 h: number analyzed (Participants) | 14 | 16 | 16 | 16
  Day 1, 8-9 h | 81.07 (15.185) | 81.41 (17.908) | 77.97 (12.859) | 82.38 (11.944)
  Day 1, 9-10 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 9-10 h | 79.38 (16.201) | 79.31 (16.239) | 75.53 (14.272) | 82.94 (11.000)
  Day 1, 10-11 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 10-11 h | 76.54 (19.338) | 76.03 (15.206) | 72.33 (11.083) | 81.88 (10.888)
  Day 1, 11-12 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 11-12 h | 74.33 (17.192) | 74.16 (14.162) | 69.25 (10.907) | 79.76 (9.416)
  Day 1, 12-13 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 12-13 h | 74.70 (16.493) | 71.53 (16.620) | 71.16 (13.766) | 80.17 (11.182)
  Day 1, 13-14 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 13-14 h | 70.17 (16.547) | 71.00 (13.837) | 70.50 (11.540) | 79.26 (9.203)
  Day 1, 14-15 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 14-15 h | 68.47 (15.015) | 69.41 (14.053) | 70.19 (11.542) | 77.41 (7.912)
  Day 1, 15-16 h: number analyzed (Participants) | 15 | 16 | 15 | 16
  Day 1, 15-16 h | 67.30 (13.618) | 66.69 (14.791) | 68.27 (13.843) | 75.00 (8.828)
  Day 1, 16-17 h: number analyzed (Participants) | 14 | 16 | 15 | 16
  Day 1, 16-17 h | 65.75 (12.667) | 65.75 (12.031) | 67.87 (11.999) | 73.84 (8.408)
  Day 1, 17-18 h: number analyzed (Participants) | 15 | 15 | 15 | 17
  Day 1, 17-18 h | 64.20 (12.078) | 66.50 (12.102) | 65.37 (11.592) | 72.00 (8.823)
  Day 1, 18-19 h: number analyzed (Participants) | 15 | 16 | 14 | 17
  Day 1, 18-19 h | 63.34 (11.705) | 66.53 (10.848) | 67.82 (17.133) | 72.35 (6.451)
  Day 1, 19-20 h: number analyzed (Participants) | 13 | 16 | 14 | 15
  Day 1, 19-20 h | 63.58 (11.302) | 63.31 (9.889) | 70.86 (19.586) | 74.17 (11.231)
  Day 1, 20-21 h: number analyzed (Participants) | 15 | 16 | 14 | 16
  Day 1, 20-21 h | 68.81 (13.465) | 66.88 (14.906) | 70.82 (17.638) | 76.72 (11.240)
  Day 1, 21-22 h: number analyzed (Participants) | 15 | 14 | 15 | 16
  Day 1, 21-22 h | 75.23 (14.859) | 78.79 (17.327) | 71.47 (18.402) | 82.03 (13.237)
  Day 1, 22-23 h: number analyzed (Participants) | 13 | 15 | 15 | 16
  Day 1, 22-23 h | 75.08 (15.643) | 74.10 (11.235) | 70.37 (10.167) | 80.55 (13.168)
  Day 1, 23-24 h: number analyzed (Participants) | 14 | 16 | 16 | 17
  Day 1, 23-24 h | 70.21 (13.674) | 70.51 (12.439) | 69.63 (12.911) | 76.94 (12.137)
  Day 7, 0-1 h: number analyzed (Participants) | 16 | 15 | 12 | 13
  Day 7, 0-1 h | 73.97 (12.115) | 68.25 (12.667) | 69.79 (10.700) | 75.07 (13.723)
  Day 7, 1-2 h: number analyzed (Participants) | 14 | 15 | 13 | 13
  Day 7, 1-2 h | 76.66 (16.264) | 70.17 (13.754) | 72.63 (12.989) | 74.05 (12.343)
  Day 7, 2-3 h: number analyzed (Participants) | 14 | 13 | 14 | 12
  Day 7, 2-3 h | 74.21 (16.735) | 65.96 (13.524) | 69.89 (14.077) | 76.96 (14.353)
  Day 7, 3-4 h: number analyzed (Participants) | 15 | 13 | 14 | 14
  Day 7, 3-4 h | 75.30 (15.794) | 71.35 (16.210) | 69.30 (11.496) | 77.71 (14.097)
  Day 7, 4-5 h: number analyzed (Participants) | 13 | 12 | 12 | 12
  Day 7, 4-5 h | 83.21 (12.349) | 80.61 (14.581) | 78.96 (12.857) | 85.25 (16.055)
  Day 7, 5-6 h: number analyzed (Participants) | 15 | 14 | 14 | 13
  Day 7, 5-6 h | 90.63 (11.828) | 79.65 (17.860) | 79.12 (15.687) | 86.54 (15.224)
  Day 7, 6-7 h: number analyzed (Participants) | 15 | 14 | 14 | 13
  Day 7, 6-7 h | 90.50 (17.096) | 78.07 (13.867) | 74.69 (14.010) | 81.28 (11.328)
  Day 7, 7-8 h: number analyzed (Participants) | 14 | 15 | 13 | 13
  Day 7, 7-8 h | 90.93 (16.769) | 74.63 (12.662) | 74.56 (13.507) | 81.15 (13.423)
  Day 7, 8-9 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 8-9 h | 85.50 (12.923) | 76.53 (14.341) | 76.40 (14.970) | 81.57 (15.587)
  Day 7, 9-10 h: number analyzed (Participants) | 15 | 15 | 13 | 13
  Day 7, 9-10 h | 78.60 (12.900) | 75.73 (14.007) | 76.88 (12.395) | 88.00 (14.735)
  Day 7, 10-11 h: number analyzed (Participants) | 15 | 15 | 14 | 14
  Day 7, 10-11 h | 78.80 (12.846) | 75.83 (15.496) | 79.63 (15.493) | 82.17 (12.757)
  Day 7, 11-12 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 11-12 h | 77.17 (12.349) | 73.61 (12.435) | 75.55 (13.549) | 82.03 (9.553)
  Day 7, 12-13 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 12-13 h | 74.47 (16.722) | 72.23 (13.522) | 75.23 (12.760) | 81.47 (9.021)
  Day 7, 13-14 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 13-14 h | 73.90 (16.245) | 70.10 (13.925) | 73.26 (13.101) | 80.37 (8.423)
  Day 7, 14-15 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 14-15 h | 67.97 (14.851) | 70.10 (13.288) | 72.50 (11.970) | 80.37 (8.943)
  Day 7, 15-16 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 15-16 h | 69.00 (14.210) | 66.70 (11.188) | 71.98 (10.818) | 75.80 (8.988)
  Day 7, 16-17 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 16-17 h | 66.47 (13.970) | 65.60 (10.524) | 70.83 (10.822) | 74.73 (9.243)
  Day 7, 17-18 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 17-18 h | 66.60 (13.494) | 65.57 (10.962) | 70.75 (12.194) | 74.23 (8.542)
  Day 7, 18-19 h: number analyzed (Participants) | 15 | 14 | 14 | 15
  Day 7, 18-19 h | 65.27 (14.732) | 66.64 (9.976) | 69.07 (10.887) | 74.10 (10.369)
  Day 7, 19-20 h: number analyzed (Participants) | 14 | 14 | 14 | 15
  Day 7, 19-20 h | 67.89 (15.134) | 67.17 (11.047) | 68.86 (13.388) | 73.47 (9.066)
  Day 7, 20-21 h: number analyzed (Participants) | 14 | 13 | 14 | 13
  Day 7, 20-21 h | 69.75 (15.978) | 67.35 (15.498) | 68.39 (14.531) | 75.12 (13.670)
  Day 7, 21-22 h: number analyzed (Participants) | 14 | 14 | 14 | 15
  Day 7, 21-22 h | 81.25 (17.242) | 70.39 (14.987) | 75.08 (18.779) | 81.10 (18.165)
  Day 7, 22-23 h: number analyzed (Participants) | 15 | 13 | 14 | 14
  Day 7, 22-23 h | 78.27 (17.026) | 71.85 (22.724) | 72.96 (13.181) | 83.00 (16.501)
  Day 7, 23-24 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 23-24 h | 73.90 (16.937) | 69.51 (10.521) | 71.79 (12.076) | 76.50 (12.890)
  Day 14, 0-1 h: number analyzed (Participants) | 15 | 14 | 12 | 14
  Day 14, 0-1 h | 72.58 (13.911) | 69.26 (12.264) | 71.43 (12.365) | 71.31 (11.094)
  Day 14, 1-2 h: number analyzed (Participants) | 15 | 13 | 11 | 13
  Day 14, 1-2 h | 70.73 (12.767) | 67.31 (10.363) | 73.09 (14.935) | 79.42 (14.377)
  Day 14, 2-3 h: number analyzed (Participants) | 15 | 13 | 12 | 12
  Day 14, 2-3 h | 69.30 (15.013) | 69.00 (13.952) | 73.79 (15.563) | 80.38 (11.531)
  Day 14, 3-4 h: number analyzed (Participants) | 16 | 15 | 12 | 11
  Day 14, 3-4 h | 74.81 (16.120) | 69.70 (11.730) | 72.72 (11.496) | 77.95 (10.489)
  Day 14, 4-5 h: number analyzed (Participants) | 16 | 15 | 11 | 13
  Day 14, 4-5 h | 83.09 (18.120) | 76.30 (15.787) | 77.08 (12.802) | 81.46 (13.089)
  Day 14, 5-6 h: number analyzed (Participants) | 15 | 15 | 11 | 13
  Day 14, 5-6 h | 87.17 (13.308) | 76.63 (13.348) | 81.53 (11.850) | 89.15 (14.899)
  Day 14, 6-7 h: number analyzed (Participants) | 14 | 13 | 12 | 12
  Day 14, 6-7 h | 81.62 (11.162) | 75.29 (12.525) | 77.92 (15.697) | 87.79 (16.734)
  Day 14, 7-8 h: number analyzed (Participants) | 15 | 15 | 11 | 13
  Day 14, 7-8 h | 79.77 (14.674) | 77.10 (15.826) | 76.32 (15.363) | 77.67 (13.774)
  Day 14, 8-9 h: number analyzed (Participants) | 16 | 15 | 13 | 12
  Day 14, 8-9 h | 79.97 (13.840) | 77.03 (13.345) | 76.77 (12.882) | 81.17 (10.069)
  Day 14, 9-10 h: number analyzed (Participants) | 16 | 14 | 13 | 14
  Day 14, 9-10 h | 77.38 (14.157) | 80.21 (18.824) | 77.65 (16.831) | 82.89 (7.669)
  Day 14, 10-11 h: number analyzed (Participants) | 14 | 15 | 13 | 14
  Day 14, 10-11 h | 81.14 (11.396) | 74.27 (15.734) | 78.85 (18.580) | 80.71 (7.844)
  Day 14, 11-12 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 11-12 h | 78.78 (12.658) | 74.60 (11.558) | 76.65 (14.867) | 79.75 (8.512)
  Day 14, 12-13 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 12-13 h | 76.53 (12.925) | 71.40 (14.023) | 73.85 (12.556) | 80.54 (8.434)
  Day 14, 13-14 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 13-14 h | 74.09 (13.790) | 71.33 (13.282) | 74.96 (14.060) | 77.43 (8.216)
  Day 14, 14-15 h: number analyzed (Participants) | 16 | 15 | 12 | 14
  Day 14, 14-15 h | 71.41 (14.672) | 69.73 (11.654) | 74.78 (13.677) | 78.18 (10.622)
  Day 14, 15-16 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 15-16 h | 70.72 (12.920) | 68.87 (12.238) | 71.62 (12.805) | 76.21 (7.300)
  Day 14, 16-17 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 16-17 h | 69.16 (11.226) | 65.10 (11.382) | 73.65 (11.067) | 74.79 (8.937)
  Day 14, 17-18 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 17-18 h | 69.53 (12.929) | 63.87 (12.354) | 72.96 (11.684) | 72.46 (8.439)
  Day 14, 18-19 h: number analyzed (Participants) | 16 | 15 | 12 | 14
  Day 14, 18-19 h | 66.72 (10.807) | 64.60 (12.689) | 69.83 (12.394) | 71.43 (8.408)
  Day 14, 19-20 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 19-20 h | 66.25 (11.703) | 65.33 (13.591) | 67.59 (11.334) | 72.04 (8.734)
  Day 14, 20-21 h: number analyzed (Participants) | 16 | 13 | 12 | 12
  Day 14, 20-21 h | 72.56 (16.361) | 68.31 (16.095) | 71.17 (15.336) | 70.63 (9.163)
  Day 14, 21-22 h: number analyzed (Participants) | 15 | 15 | 13 | 13
  Day 14, 21-22 h | 79.67 (17.424) | 70.73 (13.157) | 79.31 (17.590) | 77.92 (12.715)
  Day 14, 22-23 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 22-23 h | 77.15 (14.389) | 71.67 (14.608) | 75.58 (10.004) | 78.46 (9.268)
  Day 14, 23-24 h: number analyzed (Participants) | 16 | 14 | 13 | 14
  Day 14, 23-24 h | 79.06 (16.986) | 67.82 (11.478) | 70.23 (10.633) | 78.39 (16.352)

8. Secondary Outcome: Mean Maximum Hourly HR 0-24 h at Day 1, 7 and 14
Description: HR was measured using 28.5 h ABPM. The assessments for maximum HR were analyzed hourly as 0-1 h, 1-2 h, 2-3 h, 3-4 h, 4-5 h, 5-6 h, 6-7 h, 7-8 h, 8-9 h, 9-10 h, 10-11 h, 11-12 h, 12-13 h, 13-14 h, 14-15 h, 15-16 h, 16-17 h, 17-18 h, 18-19 h, 19-20 h, 20-21 h, 21-22 h, 22-23 h and 23-24 h at Day 1, Day 7 and Day 14.
Time Frame: Day 1 up to Day 14
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
bpm
  Day 1, 0-1 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 0-1 h | 70.6 (13.01) | 71.1 (12.33) | 74.4 (15.08) | 76.6 (10.98)
  Day 1, 1-2 h: number analyzed (Participants) | 15 | 16 | 15 | 17
  Day 1, 1-2 h | 72.2 (15.32) | 72.8 (16.72) | 76.4 (16.21) | 74.1 (10.19)
  Day 1, 2-3 h: number analyzed (Participants) | 15 | 12 | 16 | 14
  Day 1, 2-3 h | 75.8 (19.33) | 70.1 (17.21) | 71.8 (17.31) | 78.6 (12.08)
  Day 1, 3-4 h: number analyzed (Participants) | 13 | 15 | 15 | 16
  Day 1, 3-4 h | 71.2 (14.27) | 74.4 (15.90) | 72.8 (12.69) | 78.2 (11.11)
  Day 1, 4-5 h: number analyzed (Participants) | 14 | 16 | 16 | 16
  Day 1, 4-5 h | 84.6 (22.67) | 78.0 (18.81) | 81.6 (14.40) | 86.4 (12.91)
  Day 1, 5-6 h: number analyzed (Participants) | 14 | 14 | 15 | 15
  Day 1, 5-6 h | 94.2 (18.14) | 82.3 (16.45) | 86.4 (11.38) | 88.5 (18.88)
  Day 1, 6-7 h: number analyzed (Participants) | 14 | 15 | 16 | 14
  Day 1, 6-7 h | 89.6 (18.90) | 80.5 (17.73) | 78.9 (13.44) | 83.1 (12.07)
  Day 1, 7-8 h: number analyzed (Participants) | 12 | 16 | 15 | 15
  Day 1, 7-8 h | 84.9 (17.74) | 84.5 (19.89) | 80.2 (16.38) | 84.4 (13.92)
  Day 1, 8-9 h: number analyzed (Participants) | 14 | 16 | 16 | 16
  Day 1, 8-9 h | 85.0 (17.26) | 84.2 (19.19) | 81.1 (13.49) | 85.1 (13.11)
  Day 1, 9-10 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 9-10 h | 82.4 (15.48) | 82.2 (15.71) | 77.3 (14.85) | 84.6 (11.70)
  Day 1, 10-11 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 10-11 h | 78.7 (19.80) | 78.9 (17.02) | 74.1 (11.79) | 84.4 (12.47)
  Day 1, 11-12 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 11-12 h | 75.9 (17.39) | 75.9 (14.90) | 71.3 (12.00) | 82.0 (9.87)
  Day 1, 12-13 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 12-13 h | 77.3 (17.59) | 73.4 (17.79) | 74.3 (17.66) | 83.0 (12.34)
  Day 1, 13-14 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 13-14 h | 71.5 (16.84) | 72.4 (14.33) | 72.7 (12.04) | 81.4 (10.35)
  Day 1, 14-15 h: number analyzed (Participants) | 15 | 16 | 16 | 17
  Day 1, 14-15 h | 69.7 (14.69) | 70.8 (14.61) | 71.8 (12.41) | 79.8 (7.82)
  Day 1, 15-16 h: number analyzed (Participants) | 15 | 16 | 15 | 16
  Day 1, 15-16 h | 68.9 (13.69) | 68.9 (17.61) | 69.2 (13.96) | 76.1 (8.84)
  Day 1, 16-17 h: number analyzed (Participants) | 14 | 16 | 15 | 16
  Day 1, 16-17 h | 68.1 (13.32) | 67.6 (12.10) | 70.9 (13.24) | 76.2 (9.06)
  Day 1, 17-18 h: number analyzed (Participants) | 15 | 15 | 15 | 17
  Day 1, 17-18 h | 65.6 (11.67) | 68.9 (13.30) | 67.0 (11.47) | 74.2 (9.28)
  Day 1, 18-19 h: number analyzed (Participants) | 15 | 16 | 14 | 17
  Day 1, 18-19 h | 64.9 (11.94) | 70.9 (13.15) | 70.4 (17.35) | 75.7 (7.54)
  Day 1, 19-20 h: number analyzed (Participants) | 13 | 16 | 14 | 15
  Day 1, 19-20 h | 65.5 (12.14) | 64.7 (10.82) | 73.8 (19.57) | 77.2 (13.61)
  Day 1, 20-21 h: number analyzed (Participants) | 15 | 16 | 14 | 16
  Day 1, 20-21 h | 71.7 (14.17) | 71.3 (17.68) | 72.6 (18.91) | 79.9 (12.54)
  Day 1, 21-22 h: number analyzed (Participants) | 15 | 14 | 15 | 16
  Day 1, 21-22 h | 77.6 (15.88) | 85.0 (25.45) | 72.7 (19.60) | 84.3 (14.31)
  Day 1, 22-23 h: number analyzed (Participants) | 13 | 15 | 15 | 16
  Day 1, 22-23 h | 77.1 (15.50) | 79.5 (15.12) | 71.9 (10.79) | 82.9 (14.73)
  Day 1, 23-24 h: number analyzed (Participants) | 14 | 16 | 16 | 17
  Day 1, 23-24 h | 72.6 (12.87) | 72.1 (12.83) | 71.7 (12.59) | 79.1 (12.78)
  Day 7, 0-1 h: number analyzed (Participants) | 16 | 15 | 12 | 13
  Day 7, 0-1 h | 78.4 (12.21) | 71.4 (13.82) | 73.2 (12.13) | 77.2 (14.04)
  Day 7, 1-2 h: number analyzed (Participants) | 14 | 15 | 13 | 13
  Day 7, 1-2 h | 78.9 (16.88) | 73.0 (15.46) | 75.5 (13.53) | 74.8 (12.30)
  Day 7, 2-3 h: number analyzed (Participants) | 14 | 13 | 14 | 12
  Day 7, 2-3 h | 75.5 (16.70) | 67.2 (13.83) | 71.4 (14.32) | 77.9 (14.93)
  Day 7, 3-4 h: number analyzed (Participants) | 15 | 13 | 14 | 14
  Day 7, 3-4 h | 77.5 (15.32) | 73.3 (17.38) | 71.0 (11.78) | 80.0 (14.22)
  Day 7, 4-5 h: number analyzed (Participants) | 13 | 12 | 12 | 12
  Day 7, 4-5 h | 88.8 (13.85) | 87.8 (18.56) | 83.1 (18.52) | 88.8 (15.42)
  Day 7, 5-6 h: number analyzed (Participants) | 15 | 14 | 14 | 13
  Day 7, 5-6 h | 94.0 (13.05) | 82.1 (17.81) | 80.7 (16.52) | 88.8 (16.11)
  Day 7, 6-7 h: number analyzed (Participants) | 15 | 14 | 14 | 13
  Day 7, 6-7 h | 92.5 (16.78) | 85.4 (15.58) | 76.6 (13.91) | 83.8 (12.81)
  Day 7, 7-8 h: number analyzed (Participants) | 14 | 15 | 13 | 13
  Day 7, 7-8 h | 96.7 (20.74) | 77.9 (13.02) | 77.6 (16.31) | 83.9 (14.41)
  Day 7, 8-9 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 8-9 h | 89.2 (12.96) | 78.5 (15.27) | 77.8 (15.41) | 84.1 (17.28)
  Day 7, 9-10 h: number analyzed (Participants) | 15 | 15 | 13 | 13
  Day 7, 9-10 h | 81.9 (14.09) | 77.5 (13.84) | 80.0 (13.27) | 91.2 (16.05)
  Day 7, 10-11 h: number analyzed (Participants) | 15 | 15 | 14 | 14
  Day 7, 10-11 h | 83.2 (13.12) | 78.5 (17.13) | 83.1 (16.04) | 84.6 (13.56)
  Day 7, 11-12 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 11-12 h | 81.2 (12.64) | 75.3 (12.58) | 77.2 (14.04) | 83.6 (9.63)
  Day 7, 12-13 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 12-13 h | 77.2 (17.63) | 74.5 (13.51) | 77.3 (13.33) | 83.4 (8.86)
  Day 7, 13-14 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 13-14 h | 76.5 (16.76) | 71.7 (14.67) | 75.6 (14.16) | 82.1 (9.38)
  Day 7, 14-15 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 14-15 h | 69.4 (15.55) | 72.6 (13.56) | 74.4 (12.64) | 83.2 (10.35)
  Day 7, 15-16 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 15-16 h | 71.3 (15.41) | 68.5 (11.80) | 74.0 (11.31) | 77.1 (8.83)
  Day 7, 16-17 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 16-17 h | 68.3 (15.42) | 67.3 (11.30) | 73.4 (11.95) | 76.7 (8.67)
  Day 7, 17-18 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 17-18 h | 68.9 (14.09) | 67.1 (11.08) | 72.7 (13.78) | 75.7 (9.43)
  Day 7, 18-19 h: number analyzed (Participants) | 15 | 14 | 14 | 15
  Day 7, 18-19 h | 66.3 (14.80) | 68.9 (9.86) | 72.5 (12.40) | 76.3 (11.03)
  Day 7, 19-20 h: number analyzed (Participants) | 14 | 14 | 14 | 15
  Day 7, 19-20 h | 71.7 (18.46) | 69.9 (12.47) | 71.2 (13.45) | 75.3 (9.36)
  Day 7, 20-21 h: number analyzed (Participants) | 14 | 13 | 14 | 13
  Day 7, 20-21 h | 77.1 (16.13) | 69.6 (17.11) | 70.9 (15.08) | 76.5 (13.96)
  Day 7, 21-22 h: number analyzed (Participants) | 14 | 14 | 14 | 15
  Day 7, 21-22 h | 88.0 (20.26) | 72.0 (15.09) | 79.1 (22.11) | 83.5 (17.91)
  Day 7, 22-23 h: number analyzed (Participants) | 15 | 13 | 14 | 14
  Day 7, 22-23 h | 79.9 (18.30) | 77.2 (30.30) | 74.9 (13.45) | 86.2 (16.30)
  Day 7, 23-24 h: number analyzed (Participants) | 15 | 15 | 14 | 15
  Day 7, 23-24 h | 77.0 (17.25) | 72.1 (11.53) | 73.8 (11.45) | 78.0 (13.19)
  Day 14, 0-1 h: number analyzed (Participants) | 15 | 14 | 12 | 14
  Day 14, 0-1 h | 75.9 (15.22) | 73.1 (14.62) | 72.8 (13.24) | 74.2 (9.69)
  Day 14, 1-2 h: number analyzed (Participants) | 15 | 13 | 11 | 13
  Day 14, 1-2 h | 73.3 (12.25) | 69.8 (10.50) | 77.6 (16.51) | 81.7 (15.38)
  Day 14, 2-3 h: number analyzed (Participants) | 15 | 13 | 12 | 12
  Day 14, 2-3 h | 71.5 (15.13) | 70.8 (15.09) | 75.8 (17.29) | 81.6 (11.05)
  Day 14, 3-4 h: number analyzed (Participants) | 16 | 15 | 12 | 11
  Day 14, 3-4 h | 78.0 (17.88) | 72.9 (13.43) | 75.4 (11.35) | 79.1 (11.09)
  Day 14, 4-5 h: number analyzed (Participants) | 16 | 15 | 11 | 13
  Day 14, 4-5 h | 87.1 (16.80) | 78.6 (17.84) | 81.5 (22.85) | 83.9 (13.79)
  Day 14, 5-6 h: number analyzed (Participants) | 15 | 15 | 11 | 13
  Day 14, 5-6 h | 90.1 (13.99) | 81.1 (12.15) | 84.3 (11.71) | 91.7 (14.65)
  Day 14, 6-7 h: number analyzed (Participants) | 14 | 13 | 12 | 12
  Day 14, 6-7 h | 84.8 (9.97) | 77.8 (12.97) | 79.6 (16.19) | 88.8 (16.61)
  Day 14, 7-8 h: number analyzed (Participants) | 15 | 15 | 11 | 13
  Day 14, 7-8 h | 82.9 (14.36) | 81.5 (17.22) | 79.1 (16.53) | 80.2 (14.88)
  Day 14, 8-9 h: number analyzed (Participants) | 16 | 15 | 13 | 12
  Day 14, 8-9 h | 82.5 (14.33) | 78.6 (14.21) | 78.8 (13.74) | 82.4 (9.98)
  Day 14, 9-10 h: number analyzed (Participants) | 16 | 14 | 13 | 14
  Day 14, 9-10 h | 80.0 (15.11) | 83.6 (19.68) | 80.2 (16.58) | 85.5 (8.06)
  Day 14, 10-11 h: number analyzed (Participants) | 14 | 15 | 13 | 14
  Day 14, 10-11 h | 84.4 (11.60) | 76.3 (15.94) | 81.2 (19.62) | 82.8 (7.90)
  Day 14, 11-112 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 11-112 h | 81.6 (12.96) | 75.9 (12.31) | 78.6 (15.41) | 81.5 (8.69)
  Day 14, 12-13 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 12-13 h | 79.8 (15.21) | 74.7 (14.00) | 76.5 (13.40) | 82.6 (9.41)
  Day 14, 13-14 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 13-14 h | 76.3 (14.07) | 73.3 (14.41) | 77.1 (16.06) | 80.0 (7.62)
  Day 14, 14-15 h: number analyzed (Participants) | 16 | 15 | 12 | 14
  Day 14, 14-15 h | 73.3 (14.92) | 71.9 (11.68) | 77.1 (14.58) | 79.9 (11.16)
  Day 14, 15-16 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 15-16 h | 72.9 (13.94) | 70.7 (13.11) | 74.1 (14.21) | 78.0 (7.81)
  Day 14, 16-17 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 16-17 h | 70.8 (11.48) | 66.3 (11.78) | 76.1 (11.97) | 77.4 (10.28)
  Day 14, 17-18 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 17-18 h | 72.8 (15.25) | 65.4 (12.55) | 75.4 (12.27) | 73.8 (8.49)
  Day 14, 18-19 h: number analyzed (Participants) | 16 | 15 | 12 | 14
  Day 14, 18-19 h | 69.1 (11.03) | 67.1 (14.08) | 71.6 (12.67) | 73.5 (8.92)
  Day 14, 19-20 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 19-20 h | 68.5 (12.76) | 66.9 (14.52) | 68.8 (11.45) | 73.9 (8.53)
  Day 14, 20-21 h: number analyzed (Participants) | 16 | 13 | 12 | 12
  Day 14, 20-21 h | 75.1 (17.38) | 72.5 (20.28) | 73.3 (14.81) | 72.8 (10.21)
  Day 14, 21-22 h: number analyzed (Participants) | 15 | 15 | 13 | 13
  Day 14, 21-22 h | 82.0 (19.41) | 72.9 (13.44) | 81.8 (17.49) | 81.4 (15.05)
  Day 14, 22-23 h: number analyzed (Participants) | 16 | 15 | 13 | 14
  Day 14, 22-23 h | 79.8 (14.88) | 74.0 (14.39) | 79.8 (8.92) | 81.4 (10.13)
  Day 14, 23-24 h: number analyzed (Participants) | 16 | 14 | 13 | 14
  Day 14, 23-24 h | 81.2 (17.96) | 70.1 (11.82) | 71.5 (10.64) | 83.2 (22.59)

9. Secondary Outcome: Change From Baseline in Weighted Mean Systolic and Diastolic Blood Pressure (SBP and DBP) Derived From 28.5 h ABPM Over Time
Description: BP was measured using 28.5 h ABPM. Weighted mean SBP and DBP at 0-4 h post-dose was obtained on Day 1, 2, 7, 8, 14 and 15. Weighted mean SBP and DBP at 0-24 h post-dose was obtained on Day 1, 7 and 14. Weighted mean was calculated by calculating the AUC, and then dividing by the relevant time interval. AUC was calculated using the trapezoidal rule. Baseline was defined as the weighted mean SBP and DBP on pre-dose Day 1. The weighted mean change from Baseline was the AAUCMB. Data is reported for change from Baseline in weighted mean pre-dose values at Day 7 and Day 14; change from Baseline in weighted mean over 0-4 h at Day 1, 2, 7, 8, 14 and 15; and change from Baseline in weighted mean over 0-24 h at Day 1, 7 and 14.
Time Frame: Baseline (Day 1, pre-dose) up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
Millimeter of mercury (mmHg)
  SBP, Day 7, pre-dose: number analyzed (Participants) | 12 | 14 | 11 | 11
  SBP, Day 7, pre-dose | -7.21 (10.073) | -4.54 (16.602) | -1.67 (9.823) | -6.55 (8.572)
  SBP, Day 14, pre-dose: number analyzed (Participants) | 12 | 13 | 10 | 9
  SBP, Day 14, pre-dose | -6.17 (9.602) | -4.15 (17.991) | -1.39 (10.228) | -12.06 (14.143)
  SBP, Day 1, 0-4 h: number analyzed (Participants) | 13 | 16 | 15 | 14
  SBP, Day 1, 0-4 h | -3.99 (7.343) | -6.18 (7.152) | -3.23 (10.613) | -4.27 (8.566)
  SBP, Day 2, 0-4 h: number analyzed (Participants) | 12 | 16 | 15 | 12
  SBP, Day 2, 0-4 h | -8.96 (12.423) | -11.76 (11.715) | -5.73 (7.883) | -7.12 (8.388)
  SBP, Day 7, 0-4 h: number analyzed (Participants) | 12 | 14 | 11 | 11
  SBP, Day 7, 0-4 h | -8.98 (9.838) | -7.86 (10.724) | -2.43 (8.855) | -8.34 (11.266)
  SBP, Day 8, 0-4 h: number analyzed (Participants) | 12 | 14 | 12 | 11
  SBP, Day 8, 0-4 h | -11.11 (11.261) | -10.67 (10.713) | -6.14 (14.561) | -13.42 (13.907)
  SBP, Day 14, 0-4 h: number analyzed (Participants) | 12 | 13 | 10 | 9
  SBP, Day 14, 0-4 h | -8.82 (12.338) | -8.14 (9.324) | -9.36 (10.142) | -11.06 (13.844)
  SBP, Day 15, 0-4 h: number analyzed (Participants) | 12 | 14 | 10 | 11
  SBP, Day 15, 0-4 h | -7.96 (9.639) | -11.86 (13.264) | -11.27 (11.249) | -14.97 (11.794)
  SBP, Day 7, 0-24 h: number analyzed (Participants) | 12 | 14 | 11 | 11
  SBP, Day 7, 0-24 h | -13.76 (10.592) | -15.34 (11.591) | -7.75 (7.552) | -14.82 (10.810)
  SBP, Day 14, 0-24 h: number analyzed (Participants) | 12 | 13 | 10 | 9
  SBP, Day 14, 0-24 h | -14.29 (12.265) | -14.13 (11.422) | -12.79 (10.319) | -14.34 (10.636)
  DBP, Day 7, pre-dose: number analyzed (Participants) | 12 | 14 | 11 | 11
  DBP, Day 7, pre-dose | -0.60 (8.011) | 0.21 (9.021) | -0.33 (5.888) | -5.59 (7.151)
  DBP, Day 14, pre-dose: number analyzed (Participants) | 12 | 13 | 10 | 9
  DBP, Day 14, pre-dose | -0.71 (7.733) | -0.88 (8.530) | -0.17 (8.108) | -6.89 (9.168)
  DBP, Day 1, 0-4 h: number analyzed (Participants) | 13 | 16 | 15 | 14
  DBP, Day 1, 0-4 h | 2.72 (5.654) | -1.49 (5.611) | 0.95 (7.894) | -5.04 (4.220)
  DBP, Day 2, 0-4 h: number analyzed (Participants) | 12 | 16 | 15 | 12
  DBP, Day 2, 0-4 h | -0.11 (5.750) | -5.02 (6.872) | -2.24 (4.980) | -5.29 (3.166)
  DBP, Day 7, 0-4 h: number analyzed (Participants) | 12 | 14 | 11 | 11
  DBP, Day 7, 0-4 h | 0.90 (6.246) | -1.39 (5.360) | -1.39 (4.325) | -7.13 (8.469)
  DBP, Day 8, 0-4 h: number analyzed (Participants) | 12 | 14 | 12 | 11
  DBP, Day 8, 0-4 h | -1.13 (7.097) | -3.64 (5.083) | -0.97 (6.468) | -10.18 (10.093)
  DBP, Day 14, 0-4 h: number analyzed (Participants) | 12 | 13 | 10 | 9
  DBP, Day 14, 0-4 h | -2.62 (7.857) | -2.89 (5.849) | -3.20 (7.134) | -7.43 (10.323)
  DBP, Day 15, 0-4 h: number analyzed (Participants) | 12 | 14 | 10 | 11
  DBP, Day 15, 0-4 h | -1.26 (4.685) | -2.78 (4.980) | -4.76 (5.665) | -9.34 (10.566)
  DBP, Day 7, 0-24 h: number analyzed (Participants) | 12 | 14 | 11 | 11
  DBP, Day 7, 0-24 h | -5.46 (7.290) | -7.28 (5.863) | -4.50 (4.737) | -13.97 (7.610)
  DBP, Day 14, 0-24 h: number analyzed (Participants) | 12 | 13 | 10 | 9
  DBP, Day 14, 0-24 h | -7.75 (7.996) | -7.95 (6.409) | -5.91 (6.979) | -12.53 (8.622)

10. Secondary Outcome: Change From Baseline in Maximum SBP and Minimum DBP Derived From 28.5 h ABPM Over Time
Description: BP was measured using 28.5 h ABPM. Maximum SBP and minimum DBP at 0-4 h post-dose was obtained on Day 1, 2, 7, 8, 14 and 15. For the calculation of 0-4 h maximum/minimum change from Baseline, measurements post-dose up to 6 h (actual time) was included. Baseline was defined as the pre-dose weighted mean of Day 1 for SBP and DBP. Maximum/minimum change from Baseline was calculated by subtracting the Baseline value (weighted mean pre-dose Day 1 for SBP and DBP) from the maximum/minimum assessment value (during 0-4 h) of the individual post-Baseline time points.
Time Frame: Baseline (Day 1, pre-dose) up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
mmHg
  Maximum SBP, Day 1: number analyzed (Participants) | 14 | 16 | 15 | 15
  Maximum SBP, Day 1 | 11.2 (9.46) | 11.8 (6.77) | 14.5 (11.26) | 9.3 (9.56)
  Maximum SBP, Day 2: number analyzed (Participants) | 12 | 16 | 15 | 14
  Maximum SBP, Day 2 | 2.8 (14.31) | 2.8 (12.34) | 10.2 (11.49) | 4.4 (9.38)
  Maximum SBP, Day 7: number analyzed (Participants) | 13 | 15 | 12 | 11
  Maximum SBP, Day 7 | 6.9 (10.06) | 8.8 (13.91) | 14.5 (8.55) | 2.8 (13.80)
  Maximum SBP, Day 8: number analyzed (Participants) | 13 | 15 | 12 | 11
  Maximum SBP, Day 8 | 2.1 (11.92) | 4.2 (15.20) | 7.2 (17.17) | -1.2 (16.82)
  Maximum SBP, Day 14: number analyzed (Participants) | 13 | 15 | 10 | 11
  Maximum SBP, Day 14 | 9.1 (10.25) | 9.4 (12.89) | 8.1 (9.44) | 2.9 (14.52)
  Maximum SBP, Day 15: number analyzed (Participants) | 13 | 15 | 11 | 11
  Maximum SBP, Day 15 | 5.7 (15.38) | -2.5 (13.39) | 3.3 (12.11) | -3.3 (12.07)
  Minimum, DBP, Day 1: number analyzed (Participants) | 14 | 16 | 15 | 15
  Minimum, DBP, Day 1 | -8.3 (5.79) | -12.7 (7.93) | -11.5 (9.07) | -14.5 (4.88)
  Minimum, DBP, Day 2: number analyzed (Participants) | 12 | 16 | 15 | 14
  Minimum, DBP, Day 2 | -8.8 (7.83) | -14.0 (9.59) | -12.5 (7.21) | -15.0 (5.19)
  Minimum, DBP, Day 7: number analyzed (Participants) | 13 | 15 | 12 | 11
  Minimum, DBP, Day 7 | -9.3 (7.84) | -15.4 (9.69) | -12.2 (8.60) | -14.7 (9.33)
  Minimum, DBP, Day 8: number analyzed (Participants) | 13 | 15 | 12 | 11
  Minimum, DBP, Day 8 | -8.0 (9.67) | -13.4 (9.22) | -10.4 (8.31) | -19.2 (11.90)
  Minimum, DBP, Day 14: number analyzed (Participants) | 13 | 15 | 10 | 11
  Minimum, DBP, Day 14 | -17.0 (12.93) | -15.8 (9.62) | -16.5 (12.85) | -14.3 (10.72)
  Minimum, DBP, Day 15: number analyzed (Participants) | 13 | 15 | 11 | 11
  Minimum, DBP, Day 15 | -10.2 (6.95) | -12.2 (7.13) | -14.3 (12.37) | -17.3 (12.12)

11. Secondary Outcome: Mean Weighted Mean SBP and DBP at 0-4 h, Weighted Mean SBP and DBP at 0-24 h and Maximum SBP and Minimum DBP at 0-4 h Derived From 28.5 h ABPM
Description: BP was measured using 28.5 h ABPM. Weighted mean SBP and DBP at 0-4 h post-dose was obtained on Day 1, 2, 7, 8, 14 and 15. Weighted mean SBP and DBP at 0-24 h post-dose was obtained on Day 1, 7 and 14. Maximum SBP and minimum DBP at 0-4 h post-dose was obtained on Day 1, 2, 7, 8, 14 and 15. Baseline was defined as the pre-dose weighted mean of Day 1.
Time Frame: Day 1 up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
mmHg
  Weighted mean SBP 0-4, Day 1: number analyzed (Participants) | 13 | 16 | 15 | 14
  Weighted mean SBP 0-4, Day 1 | 130.55 (15.052) | 128.47 (11.670) | 130.66 (16.508) | 126.05 (14.111)
  Weighted mean SBP 0-4, Day 2: number analyzed (Participants) | 13 | 16 | 17 | 15
  Weighted mean SBP 0-4, Day 2 | 128.15 (18.616) | 122.90 (13.129) | 129.23 (16.139) | 124.03 (16.147)
  Weighted mean SBP 0-4, Day 7: number analyzed (Participants) | 14 | 14 | 13 | 13
  Weighted mean SBP 0-4, Day 7 | 129.32 (16.655) | 126.46 (15.897) | 130.52 (13.432) | 123.10 (12.523)
  Weighted mean SBP 0-4, Day 8: number analyzed (Participants) | 14 | 14 | 14 | 14
  Weighted mean SBP 0-4, Day 8 | 128.54 (16.817) | 123.65 (15.120) | 127.55 (13.141) | 117.26 (11.281)
  Weighted mean SBP 0-4, Day 14: number analyzed (Participants) | 15 | 13 | 11 | 12
  Weighted mean SBP 0-4, Day 14 | 130.71 (17.527) | 124.59 (9.640) | 124.86 (13.833) | 122.94 (11.670)
  Weighted mean SBP 0-4, Day 15: number analyzed (Participants) | 15 | 14 | 12 | 14
  Weighted mean SBP 0-4, Day 15 | 128.84 (17.647) | 120.74 (14.472) | 124.68 (14.886) | 118.52 (14.773)
  Weighted mean SBP 0-24, Day 1: number analyzed (Participants) | 13 | 16 | 15 | 14
  Weighted mean SBP 0-24, Day 1 | 122.64 (16.675) | 117.48 (11.246) | 124.41 (13.961) | 117.94 (11.565)
  Weighted mean SBP 0-24, Day 7: number analyzed (Participants) | 14 | 14 | 13 | 13
  Weighted mean SBP 0-24, Day 7 | 124.22 (16.893) | 118.98 (11.587) | 124.60 (12.774) | 116.34 (11.150)
  Weighted mean SBP 0-24, Day 14: number analyzed (Participants) | 15 | 13 | 11 | 12
  Weighted mean SBP 0-24, Day 14 | 125.45 (16.546) | 118.60 (8.748) | 122.71 (16.117) | 119.11 (9.109)
  Maximum SBP 0-4 h, Day 1: number analyzed (Participants) | 16 | 16 | 17 | 18
  Maximum SBP 0-4 h, Day 1 | 150.0 (18.72) | 146.4 (15.61) | 147.6 (18.78) | 141.3 (15.03)
  Maximum SBP 0-4 h, Day 2: number analyzed (Participants) | 14 | 16 | 17 | 17
  Maximum SBP 0-4 h, Day 2 | 140.0 (19.98) | 137.4 (15.78) | 145.9 (21.48) | 136.0 (16.71)
  Maximum SBP 0-4 h, Day 7: number analyzed (Participants) | 16 | 15 | 14 | 14
  Maximum SBP 0-4 h, Day 7 | 143.9 (20.10) | 142.7 (20.02) | 148.4 (18.60) | 135.5 (15.97)
  Maximum SBP 0-4 h, Day 8: number analyzed (Participants) | 15 | 15 | 14 | 14
  Maximum SBP 0-4 h, Day 8 | 141.1 (17.13) | 138.1 (19.26) | 141.8 (17.64) | 129.4 (14.06)
  Maximum SBP 0-4 h, Day 14: number analyzed (Participants) | 16 | 15 | 12 | 14
  Maximum SBP 0-4 h, Day 14 | 148.4 (20.04) | 143.3 (14.06) | 141.3 (14.43) | 135.1 (12.94)
  Maximum SBP 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 13 | 14
  Maximum SBP 0-4 h, Day 15 | 142.8 (21.83) | 131.4 (16.91) | 138.4 (13.08) | 129.8 (15.02)
  Weighted mean DBP 0-4, Day 1: number analyzed (Participants) | 13 | 16 | 15 | 14
  Weighted mean DBP 0-4, Day 1 | 82.48 (9.817) | 77.54 (8.200) | 77.46 (11.603) | 78.14 (10.879)
  Weighted mean DBP 0-4, Day 2: number analyzed (Participants) | 13 | 16 | 17 | 15
  Weighted mean DBP 0-4, Day 2 | 80.81 (9.182) | 74.01 (7.959) | 74.67 (12.607) | 77.07 (12.058)
  Weighted mean DBP 0-4, Day 7: number analyzed (Participants) | 14 | 14 | 13 | 13
  Weighted mean DBP 0-4, Day 7 | 82.83 (10.367) | 78.07 (8.744) | 74.87 (11.216) | 74.63 (8.888)
  Weighted mean DBP 0-4, Day 8: number analyzed (Participants) | 14 | 14 | 14 | 14
  Weighted mean DBP 0-4, Day 8 | 81.88 (11.151) | 75.82 (9.090) | 74.77 (10.137) | 71.24 (10.305)
  Weighted mean DBP 0-4, Day 14: number analyzed (Participants) | 15 | 13 | 11 | 12
  Weighted mean DBP 0-4, Day 14 | 81.49 (10.037) | 76.31 (4.101) | 72.14 (10.218) | 76.10 (8.595)
  Weighted mean DBP 0-4, Day 15: number analyzed (Participants) | 15 | 14 | 12 | 14
  Weighted mean DBP 0-4, Day 15 | 79.25 (9.154) | 75.25 (7.330) | 71.94 (11.908) | 73.61 (12.810)
  Weighted mean DBP 0-24, Day 1: number analyzed (Participants) | 13 | 16 | 15 | 14
  Weighted mean DBP 0-24, Day 1 | 74.44 (8.758) | 70.53 (7.941) | 71.58 (10.670) | 70.49 (10.530)
  Weighted mean DBP 0-24, Day 7: number analyzed (Participants) | 14 | 14 | 13 | 13
  Weighted mean DBP 0-24, Day 7 | 76.20 (9.831) | 72.18 (6.598) | 71.10 (10.471) | 67.46 (7.075)
  Weighted mean DBP 0-24, Day 14: number analyzed (Participants) | 15 | 13 | 11 | 12
  Weighted mean DBP 0-24, Day 14 | 76.07 (9.443) | 71.24 (5.775) | 69.95 (11.156) | 71.00 (7.793)
  Minimum DBP 0-4 h, Day 1: number analyzed (Participants) | 16 | 16 | 17 | 18
  Minimum DBP 0-4 h, Day 1 | 73.1 (9.14) | 66.4 (9.73) | 65.4 (12.03) | 69.3 (9.99)
  Minimum DBP 0-4 h, Day 2: number analyzed (Participants) | 14 | 16 | 17 | 17
  Minimum DBP 0-4 h, Day 2 | 73.6 (11.43) | 65.1 (9.74) | 63.4 (12.27) | 68.1 (12.84)
  Minimum DBP 0-4 h, Day 7: number analyzed (Participants) | 16 | 15 | 14 | 14
  Minimum DBP 0-4 h, Day 7 | 72.6 (10.55) | 63.3 (12.12) | 63.9 (11.53) | 67.1 (8.07)
  Minimum DBP 0-4 h, Day 8: number analyzed (Participants) | 15 | 15 | 14 | 14
  Minimum DBP 0-4 h, Day 8 | 74.1 (10.49) | 65.2 (11.95) | 65.1 (11.10) | 62.6 (12.38)
  Minimum DBP 0-4 h, Day 14: number analyzed (Participants) | 16 | 15 | 12 | 14
  Minimum DBP 0-4 h, Day 14 | 65.8 (14.53) | 62.8 (7.75) | 59.3 (13.32) | 67.4 (10.67)
  Minimum DBP 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 13 | 14
  Minimum DBP 0-4 h, Day 15 | 70.6 (9.17) | 66.4 (8.60) | 64.0 (15.06) | 65.6 (13.92)

12. Secondary Outcome: Change From Baseline in QTc by Federicia's Method (F) and QTc Bazett's Method (B) Values at Pre-dose, Weighted Mean 0-4 h and Maximum 0-4 h Derived From 12-lead Electrocardiogram (ECG) Over Time
Description: A 12-lead ECG was recorded on Day 1, 2, 7, 8, 14 and 15 with the participant in a supine position having rested in that position for at least 5 min before each reading. A total of 3 measurements separated by at least 1 min was taken at each visit and the mean recorded. The Baseline for pre-dose QTcF and QTcB measurements was the pre-dose assessment on Day 1. Weighted mean at 0-4 h for QTcF and QTcB was calculated by calculating the AUC, and then dividing by the relevant time interval. AUC was calculated using the trapezoidal rule. The weighted mean change from Baseline was the AAUCMB. The change from Baseline in maximum QTcF and QTcB at 0-4 h was calculated by subtracting the Baseline (pre-dose Day 1) value from the individual post-Baseline values.
Time Frame: Baseline (Day 1, pre-dose) up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millisecond (msec)
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
Millisecond (msec)
  QTcF, Day 7, pre-dose: number analyzed (Participants) | 15 | 15 | 14 | 15
  QTcF, Day 7, pre-dose | 2.548 (14.3648) | 4.166 (10.8863) | 4.557 (12.5535) | -1.622 (14.8225)
  QTcF, Day 14, pre-dose: number analyzed (Participants) | 15 | 15 | 13 | 14
  QTcF, Day 14, pre-dose | 2.445 (14.8051) | -2.215 (8.8487) | 1.450 (11.8828) | -5.803 (12.6960)
  QTcF, Weighted mean 0-4 h, Day 1: number analyzed (Participants) | 16 | 16 | 17 | 17
  QTcF, Weighted mean 0-4 h, Day 1 | 1.5102 (9.80314) | 1.2546 (7.47433) | 5.1325 (9.99564) | -0.2457 (6.77374)
  QTcF, Weighted mean 0-4 h, Day 2: number analyzed (Participants) | 16 | 16 | 17 | 16
  QTcF, Weighted mean 0-4 h, Day 2 | 1.4515 (9.95165) | 4.3733 (7.91878) | 10.5957 (16.92211) | -1.0685 (8.45786)
  QTcF, Weighted mean 0-4 h, Day 7: number analyzed (Participants) | 14 | 15 | 14 | 15
  QTcF, Weighted mean 0-4 h, Day 7 | 0.5278 (11.61138) | 3.4646 (10.28713) | 8.8287 (10.77947) | -2.6011 (14.22194)
  QTcF, Weighted mean 0-4 h, Day 8: number analyzed (Participants) | 16 | 14 | 14 | 14
  QTcF, Weighted mean 0-4 h, Day 8 | -0.2753 (13.37615) | -1.5941 (9.79215) | 8.7690 (14.91393) | -5.8609 (15.48314)
  QTcF, Weighted mean 0-4 h, Day 14: number analyzed (Participants) | 14 | 15 | 13 | 14
  QTcF, Weighted mean 0-4 h, Day 14 | 3.8254 (14.80602) | 0.8731 (8.87134) | 9.0192 (10.65315) | -3.7270 (14.27827)
  QTcF, Weighted mean 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 13 | 13
  QTcF, Weighted mean 0-4 h, Day 15 | 0.2258 (15.48959) | -2.3710 (9.06406) | 9.3434 (10.40650) | -7.9229 (9.51166)
  QTcF, Maximum 0-4 h, Day 1 | 6.138 (8.3179) | 8.099 (9.3911) | 11.169 (9.4879) | 6.334 (7.0411)
  QTcF, Maximum 0-4 h, Day 2: number analyzed (Participants) | 16 | 16 | 17 | 17
  QTcF, Maximum 0-4 h, Day 2 | 7.238 (9.8912) | 8.860 (7.1928) | 16.650 (18.1579) | 3.940 (8.4250)
  QTcF, Maximum 0-4 h, Day 7: number analyzed (Participants) | 16 | 15 | 14 | 15
  QTcF, Maximum 0-4 h, Day 7 | 7.422 (10.5173) | 8.586 (11.5664) | 14.866 (11.4977) | 2.146 (13.5782)
  QTcF, Maximum 0-4 h, Day 8: number analyzed (Participants) | 16 | 15 | 14 | 14
  QTcF, Maximum 0-4 h, Day 8 | 4.765 (14.1015) | 3.434 (8.9030) | 15.425 (14.2054) | -0.707 (16.9799)
  QTcF, Maximum 0-4 h, Day 14: number analyzed (Participants) | 16 | 15 | 13 | 14
  QTcF, Maximum 0-4 h, Day 14 | 7.713 (14.0810) | 6.651 (8.6838) | 16.715 (9.8480) | -0.394 (13.4669)
  QTcF, Maximum 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 13 | 14
  QTcF, Maximum 0-4 h, Day 15 | 5.690 (15.6489) | 1.254 (7.5156) | 15.698 (11.7395) | 0.585 (13.3811)
  QTcB, Day 7, pre-dose: number analyzed (Participants) | 15 | 15 | 14 | 15
  QTcB, Day 7, pre-dose | 3.490 (14.8170) | 4.033 (11.4412) | 3.491 (17.2891) | -0.982 (18.2505)
  QTcB, Day 14, pre-dose: number analyzed (Participants) | 15 | 15 | 13 | 14
  QTcB, Day 14, pre-dose | 2.236 (18.0863) | -2.150 (12.5311) | 0.364 (13.4871) | -6.254 (14.4987)
  QTcB, Weighted mean 0-4 h, Day 1: number analyzed (Participants) | 16 | 16 | 17 | 17
  QTcB, Weighted mean 0-4 h, Day 1 | -1.4368 (10.48286) | 1.9240 (9.38964) | 7.2528 (14.91350) | 0.4135 (7.78546)
  QTcB, Weighted mean 0-4 h, Day 2: number analyzed (Participants) | 16 | 16 | 17 | 16
  QTcB, Weighted mean 0-4 h, Day 2 | -0.8322 (11.91468) | 4.5011 (12.15813) | 12.1052 (24.42441) | 0.4464 (10.89990)
  QTcB, Weighted mean 0-4 h, Day 7: number analyzed (Participants) | 14 | 15 | 14 | 15
  QTcB, Weighted mean 0-4 h, Day 7 | 0.6551 (14.84890) | 3.1554 (11.81255) | 10.6108 (16.58029) | -1.1323 (16.11649)
  QTcB, Weighted mean 0-4 h, Day 8: number analyzed (Participants) | 16 | 14 | 14 | 14
  QTcB, Weighted mean 0-4 h, Day 8 | -2.1592 (13.74186) | -2.5879 (12.83153) | 12.5741 (22.22059) | -3.9026 (16.69124)
  QTcB, Weighted mean 0-4 h, Day 14: number analyzed (Participants) | 14 | 15 | 13 | 14
  QTcB, Weighted mean 0-4 h, Day 14 | 1.5770 (16.69052) | 1.1100 (12.02700) | 11.8220 (16.58898) | -1.9538 (15.99966)
  QTcB, Weighted mean 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 13 | 13
  QTcB, Weighted mean 0-4 h, Day 15 | 0.2536 (13.32367) | -2.1912 (13.19232) | 11.8730 (19.06660) | -5.4291 (11.64105)
  QTcB, Maximum 0-4 h, Day 1 | 4.600 (9.0150) | 9.902 (12.1193) | 15.314 (12.8527) | 8.448 (9.0077)
  QTcB, Maximum 0-4 h, Day 2: number analyzed (Participants) | 16 | 16 | 17 | 17
  QTcB, Maximum 0-4 h, Day 2 | 5.130 (12.9391) | 10.797 (11.0215) | 19.846 (26.4494) | 6.038 (10.0240)
  QTcB, Maximum 0-4 h, Day 7: number analyzed (Participants) | 16 | 15 | 14 | 5
  QTcB, Maximum 0-4 h, Day 7 | 9.599 (15.2443) | 9.884 (10.8668) | 19.748 (18.6338) | 5.125 (15.1542)
  QTcB, Maximum 0-4 h, Day 8: number analyzed (Participants) | 16 | 15 | 14 | 14
  QTcB, Maximum 0-4 h, Day 8 | 4.930 (15.4632) | 3.308 (10.8675) | 22.344 (21.0882) | 2.949 (17.3141)
  QTcB, Maximum 0-4 h, Day 14: number analyzed (Participants) | 16 | 15 | 13 | 14
  QTcB, Maximum 0-4 h, Day 14 | 6.941 (16.7794) | 7.250 (12.2421) | 20.698 (14.3145) | 1.685 (15.2440)
  QTcB, Maximum 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 13 | 14
  QTcB, Maximum 0-4 h, Day 15 | 6.646 (14.1139) | 3.569 (10.9642) | 19.933 (19.5949) | 3.343 (14.0019)

13. Secondary Outcome: Mean QTcF and QTcB Values at Pre-dose, Weighted Mean 0-4 h and Maximum 0-4 h Derived From 12-lead ECG Over Time
Description: A 12-lead ECG was recorded on Day 1, 2, 7, 8, 14 and 15 with the participant in a supine position having rested in that position for at least 5 min before each reading. A total of 3 measurements separated by at least 1 min was taken at each visit and the mean recorded. The pre-dose QTcF and QTcB assessment was done at Day 1, 7 and 14. Weighted mean at 0-4 h for QTcF and QTcB at Day 1, 2, 7, 8, 14 and 15 was calculated by calculating the AUC, and then dividing by the relevant time interval. AUC was calculated using the trapezoidal rule. The maximum QTcF and QTcB at 0-4 h was obtained at Day 1, 2, 7, 8, 14 and 15.
Time Frame: Day 1 up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
msec
  QTcF, Day 1, pre-dose | 396.518 (18.9384) | 397.667 (17.9057) | 391.300 (23.3733) | 396.361 (16.7847)
  QTcF, Day 7, pre-dose: number analyzed (Participants) | 15 | 15 | 14 | 15
  QTcF, Day 7, pre-dose | 398.828 (14.5763) | 403.565 (23.5668) | 396.804 (19.9587) | 396.897 (16.8340)
  QTcF, Day 14, pre-dose: number analyzed (Participants) | 15 | 15 | 13 | 14
  QTcF, Day 14, pre-dose | 399.599 (14.8681) | 397.184 (20.8546) | 392.524 (24.7455) | 393.522 (15.5437)
  QTcF, Weighted mean 0-4 h, Day 1: number analyzed (Participants) | 16 | 16 | 17 | 17
  QTcF, Weighted mean 0-4 h, Day 1 | 399.1571 (20.93784) | 398.9213 (18.95805) | 396.4321 (23.12234) | 396.6588 (18.71828)
  QTcF, Weighted mean 0-4 h, Day 2: number analyzed (Participants) | 16 | 16 | 17 | 16
  QTcF, Weighted mean 0-4 h, Day 2 | 399.0984 (20.76430) | 402.0399 (18.98919) | 401.8953 (23.15689) | 397.3482 (17.29841)
  QTcF, Weighted mean 0-4 h, Day 7: number analyzed (Participants) | 14 | 15 | 14 | 15
  QTcF, Weighted mean 0-4 h, Day 7 | 397.6228 (13.80395) | 402.8639 (23.36556) | 401.0754 (24.39809) | 395.9180 (19.47963)
  QTcF, Weighted mean 0-4 h, Day 8: number analyzed (Participants) | 16 | 14 | 14 | 14
  QTcF, Weighted mean 0-4 h, Day 8 | 397.3716 (18.94814) | 396.6669 (19.88573) | 401.0157 (22.80350) | 393.4643 (19.93914)
  QTcF, Weighted mean 0-4 h, Day 14: number analyzed (Participants) | 14 | 15 | 13 | 14
  QTcF, Weighted mean 0-4 h, Day 14 | 399.8488 (13.18337) | 400.2724 (19.00353) | 400.0939 (20.11137) | 395.5983 (19.45327)
  QTcF, Weighted mean 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 13 | 13
  QTcF, Weighted mean 0-4 h, Day 15 | 397.8727 (16.14803) | 397.0283 (20.64521) | 400.4180 (19.18469) | 392.3686 (16.99407)
  QTcF, Maximum 0-4 h, Day 1 | 402.656 (20.3503) | 405.766 (20.3313) | 402.468 (22.2225) | 402.696 (16.6072)
  QTcF, Maximum 0-4 h, Day 2: number analyzed (Participants) | 16 | 16 | 17 | 17
  QTcF, Maximum 0-4 h, Day 2 | 404.885 (21.1074) | 406.526 (19.2241) | 407.950 (23.4527) | 400.844 (18.8346)
  QTcF, Maximum 0-4 h, Day 7: number analyzed (Participants) | 16 | 15 | 14 | 15
  QTcF, Maximum 0-4 h, Day 7 | 405.069 (16.2300) | 407.985 (24.5587) | 407.113 (24.2679) | 400.665 (18.8396)
  QTcF, Maximum 0-4 h, Day 8: number analyzed (Participants) | 16 | 15 | 14 | 14
  QTcF, Maximum 0-4 h, Day 8 | 402.412 (17.9804) | 402.833 (19.0273) | 407.671 (21.7779) | 398.618 (20.0406)
  QTcF, Maximum 0-4 h, Day 14: number analyzed (Participants) | 16 | 15 | 13 | 14
  QTcF, Maximum 0-4 h, Day 14 | 405.360 (13.6156) | 406.050 (20.5479) | 407.790 (20.6278) | 398.931 (18.9056)
  QTcF, Maximum 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 13 | 14
  QTcF, Maximum 0-4 h, Day 15 | 403.337 (16.9640) | 400.653 (18.6693) | 406.773 (19.4447) | 399.910 (17.1580)
  QTcB, Day 1, pre-dose | 405.222 (20.8892) | 402.023 (22.2404) | 396.975 (24.1244) | 406.463 (21.3658)
  QTcB, Day 7, pre-dose: number analyzed (Participants) | 15 | 15 | 14 | 15
  QTcB, Day 7, pre-dose | 407.380 (17.7924) | 408.688 (24.8189) | 401.221 (16.6437) | 409.064 (19.5591)
  QTcB, Day 14, pre-dose: number analyzed (Participants) | 15 | 15 | 13 | 14
  QTcB, Day 14, pre-dose | 409.909 (19.5835) | 402.505 (25.5206) | 398.524 (21.6747) | 403.905 (15.6393)
  QTcB, Weighted mean 0-4 h, Day 1: number analyzed (Participants) | 16 | 16 | 17 | 17
  QTcB, Weighted mean 0-4 h, Day 1 | 405.1192 (22.72290) | 403.9471 (22.10540) | 404.2282 (23.22646) | 408.8990 (21.51019)
  QTcB, Weighted mean 0-4 h, Day 2: number analyzed (Participants) | 16 | 16 | 17 | 16
  QTcB, Weighted mean 0-4 h, Day 2 | 405.7239 (21.67872) | 406.5243 (19.43633) | 409.0807 (23.78119) | 411.1034 (18.99910)
  QTcB, Weighted mean 0-4 h, Day 7: number analyzed (Participants) | 14 | 15 | 14 | 15
  QTcB, Weighted mean 0-4 h, Day 7 | 405.1001 (14.32210) | 407.8107 (24.03156) | 408.3410 (20.23969) | 408.9141 (21.56424)
  QTcB, Weighted mean 0-4 h, Day 8: number analyzed (Participants) | 16 | 14 | 14 | 14
  QTcB, Weighted mean 0-4 h, Day 8 | 404.3968 (22.29983) | 401.5862 (24.75626) | 410.3044 (20.92796) | 406.2555 (20.30000)
  QTcB, Weighted mean 0-4 h, Day 14: number analyzed (Participants) | 14 | 15 | 13 | 14
  QTcB, Weighted mean 0-4 h, Day 14 | 409.5049 (18.03324) | 405.7653 (22.29165) | 409.9818 (19.36717) | 408.2043 (20.49320)
  QTcB, Weighted mean 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 13 | 13
  QTcB, Weighted mean 0-4 h, Day 15 | 406.8096 (20.18685) | 402.4642 (25.07009) | 410.0328 (18.49302) | 406.7532 (16.53736)
  QTcB, Maximum 0-4 h, Day 1 | 409.821 (20.9888) | 411.925 (22.5302) | 412.289 (22.9219) | 414.910 (20.9889)
  QTcB, Maximum 0-4 h, Day 2: number analyzed (Participants) | 16 | 16 | 17 | 17
  QTcB, Maximum 0-4 h, Day 2 | 411.686 (21.7606) | 412.820 (20.3513) | 416.821 (24.7489) | 414.524 (21.3863)
  QTcB, Maximum 0-4 h, Day 7: number analyzed (Participants) | 16 | 15 | 14 | 15
  QTcB, Maximum 0-4 h, Day 7 | 416.155 (18.5802) | 414.540 (22.8711) | 417.478 (21.5061) | 415.172 (20.2556)
  QTcB, Maximum 0-4 h, Day 8: number analyzed (Participants) | 16 | 15 | 14 | 14
  QTcB, Maximum 0-4 h, Day 8 | 411.486 (23.2760) | 407.963 (22.5265) | 420.074 (17.7199) | 413.107 (18.3979)
  QTcB, Maximum 0-4 h, Day 14: number analyzed (Participants) | 16 | 15 | 13 | 14
  QTcB, Maximum 0-4 h, Day 14 | 413.498 (16.8864) | 411.906 (22.0750) | 418.858 (20.5848) | 411.843 (18.6525)
  QTcB, Maximum 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 13 | 14
  QTcB, Maximum 0-4 h, Day 15 | 413.202 (22.3810) | 408.224 (23.3075) | 418.093 (18.7721) | 413.501 (14.6549)

14. Secondary Outcome: Mean of Hourly Maximums QTcF and QTcB Derived From 24 h 3-lead Holter ECG Monitoring Over Time
Description: A holter monitor is a machine that continuously records the heart's electrical activity. A 3-lead holter ECG monitoring device was used. The monitor was worn for 24 h during normal activity to record the ECG intervals. The assesmment for hourly maximums QTcF and QTcB was done on Day 1, Day 7 and Day 14. For each h of holter monitoring the maximum QTcF for that h was calculated using the maximum QT and mean HR of that given h as Maximum QT divided by (60/Mean HR)^1/3. For each h of holter monitoring the maximum QTcB for that h was calculated using the maximum QT and mean HR of that given h as Maximum QT divided by (60/Mean HR)^1/2.
Time Frame: Day 1 up to Day 14
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
msec
  Day 1, QTcF: number analyzed (Participants) | 16 | 16 | 17 | 16
  Day 1, QTcF | 474.2567 (26.91319) | 470.3755 (21.52200) | 468.4990 (28.95477) | 470.6075 (20.80669)
  Day 7, QTcF: number analyzed (Participants) | 16 | 15 | 14 | 15
  Day 7, QTcF | 471.3443 (17.96397) | 470.9166 (18.10351) | 471.2125 (30.75404) | 469.7194 (17.22701)
  Day 14, QTcF: number analyzed (Participants) | 14 | 15 | 12 | 14
  Day 14, QTcF | 471.3571 (14.87705) | 478.8226 (20.29032) | 461.4473 (32.41893) | 462.4090 (18.50928)
  Day 1, QTcB: number analyzed (Participants) | 16 | 16 | 17 | 16
  Day 1, QTcB | 491.2731 (32.55948) | 486.3962 (21.76741) | 484.1421 (31.72641) | 493.5255 (21.80365)
  Day 7, QTcB: number analyzed (Participants) | 16 | 15 | 14 | 15
  Day 7, QTcB | 491.1749 (21.97287) | 486.1238 (22.36925) | 488.0985 (33.52830) | 493.4279 (19.59523)
  Day 14, QTcB: number analyzed (Participants) | 14 | 15 | 12 | 14
  Day 14, QTcB | 489.5294 (18.51699) | 494.0542 (23.18669) | 479.8827 (36.11264) | 484.5300 (16.67519)

15. Secondary Outcome: Number of Events of Supra Ventricular Ectopics, Ventricular Ectopics and Ventricular Runs Per 24 h Derived From 3-lead Holter ECG Monitoring Over Time
Description: A holter monitor is a machine that continuously records the heart's electrical activity. A 3-lead holter ECG monitoring device was used. The monitor was worn for 24 h during normal activity to record the heart's rhythm. The assessment for the events of supra ventricular ectopics, ventricular ectopics and ventricular runs per 24 h was done on Day 1, Day 7 and Day 14.
Time Frame: Day 1 up to Day 14
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Number of events
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
Number of events
  Day 1, Supra ventricular ectopics: number analyzed (Participants) | 16 | 16 | 17 | 16
  Day 1, Supra ventricular ectopics | 107.2 (259.78) | 397.3 (982.72) | 134.9 (249.35) | 61.9 (128.69)
  Day 1, Ventricular ectopics: number analyzed (Participants) | 16 | 16 | 17 | 16
  Day 1, Ventricular ectopics | 0.0 (0.00) | 0.8 (1.65) | 3.6 (10.80) | 0.3 (1.00)
  Day 1, Ventricular runs: number analyzed (Participants) | 16 | 16 | 17 | 16
  Day 1, Ventricular runs | 0.0 (0.00) | 0.2 (0.40) | 1.0 (3.16) | 0.1 (0.25)
  Day 7, Supra ventricular ectopics: number analyzed (Participants) | 16 | 15 | 14 | 15
  Day 7, Supra ventricular ectopics | 97.8 (220.23) | 321.4 (985.25) | 442.5 (900.98) | 73.0 (120.87)
  Day 7, Ventricular ectopics: number analyzed (Participants) | 16 | 15 | 14 | 15
  Day 7, Ventricular ectopics | 1.0 (4.00) | 0.2 (0.77) | 0.2 (0.80) | 0.0 (0.00)
  Day 7, Ventricular runs: number analyzed (Participants) | 16 | 15 | 14 | 15
  Day 7, Ventricular runs | 0.1 (0.25) | 0.1 (0.26) | 0.1 (0.27) | 0.0 (0.00)
  Day 14, Supra ventricular ectopics: number analyzed (Participants) | 14 | 15 | 12 | 14
  Day 14, Supra ventricular ectopics | 27.5 (42.17) | 398.1 (1005.29) | 333.5 (821.98) | 93.3 (121.83)
  Day 14, Ventricular ectopics: number analyzed (Participants) | 14 | 15 | 12 | 14
  Day 14, Ventricular ectopics | 0.5 (1.87) | 0.4 (1.55) | 0.0 (0.00) | 0.0 (0.00)
  Day 14, Ventricular runs: number analyzed (Participants) | 14 | 15 | 12 | 14
  Day 14, Ventricular runs | 0.1 (0.27) | 0.1 (0.52) | 0.0 (0.00) | 0.0 (0.00)

16. Secondary Outcome: Number of Participants With Biochemistry Abnormal Change From Baseline Values Relative to the Normal Range at Day 7 and 14
Description: The parameters of biochemistry with their normal range included: alanine amino transferase ([ALT] 0-48 international units per liter [IU/L]), albumin (32-50 gram [g]/L), alkaline phosphatase ([ALP] 20-125 IU/L), aspartate amino transferase ([AST] 0-42 IU/L), calcium (2.12-2.56 millimole [mmol]/L, chloride (95-108 mmol/L), creatine kinase ([CK] 0-235 IU/L), creatinine (44-124 micromole [µmol]/L), direct bilirubin (0-6 µmol/L), gamma glutamyl transferase ([GGT] 0-65 IU/L), glucose (3.9-6.9 mmol/L), lactate dehydrogenase ([LDH] 0-250 IU/L), potassium (3.5-5.3 mmol/L), sodium (135-146 mmol/L), total bilirubin (0-22 µmol/L), total protein (60-85 g/L), urea (2.5-9 mmol/L) and uric acid (250-510 µmol/L). The assessments were performed on Day 1, Day 7 and Day 14. Baseline was defined as the assessment done on Day 1. Only those parameters for which at least one value of abnormality (to low or to high) change from Baseline, relative to normal ranges were reported are summarized.
Time Frame: Baseline (Day 1) up to Day 14
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
Participants
  ALT, change to high, Day 7: number analyzed (Participants) | 14 | 15 | 12 | 13
  ALT, change to high, Day 7 | 0 | 0 | 0 | 1
  AST, change to high, Day 7: number analyzed (Participants) | 14 | 15 | 12 | 13
  AST, change to high, Day 7 | 1 | 0 | 0 | 1
  AST, change to high, Day 14: number analyzed (Participants) | 14 | 15 | 13 | 10
  AST, change to high, Day 14 | 0 | 0 | 0 | 1
  Calcium, change to low, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 10
  Calcium, change to low, Day 14 | 0 | 1 | 0 | 1
  Chloride, change to low, Day 7: number analyzed (Participants) | 14 | 15 | 12 | 13
  Chloride, change to low, Day 7 | 0 | 0 | 0 | 1
  Chloride, change to high, Day 7: number analyzed (Participants) | 14 | 15 | 12 | 13
  Chloride, change to high, Day 7 | 1 | 1 | 0 | 1
  Chloride, change to high, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 10
  Chloride, change to high, Day 14 | 1 | 1 | 0 | 1
  CK, change to high, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 10
  CK, change to high, Day 14 | 0 | 0 | 1 | 0
  Direct Bilirubin, change to high, Day 7: number analyzed (Participants) | 14 | 15 | 12 | 13
  Direct Bilirubin, change to high, Day 7 | 0 | 0 | 0 | 1
  GGT, change to high, Day 7: number analyzed (Participants) | 14 | 15 | 12 | 13
  GGT, change to high, Day 7 | 0 | 1 | 0 | 1
  GGT, change to high, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 10
  GGT, change to high, Day 14 | 0 | 1 | 0 | 2
  Glucose, change to high, Day 7: number analyzed (Participants) | 14 | 15 | 12 | 13
  Glucose, change to high, Day 7 | 0 | 2 | 1 | 1
  Glucose, change to low, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 10
  Glucose, change to low, Day 14 | 0 | 0 | 0 | 1
  Glucose, change to high, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 10
  Glucose, change to high, Day 14 | 1 | 1 | 2 | 1
  LDH, change to high, Day 7: number analyzed (Participants) | 14 | 15 | 12 | 13
  LDH, change to high, Day 7 | 0 | 0 | 0 | 1
  LDH, change to high, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 10
  LDH, change to high, Day 14 | 1 | 1 | 0 | 0
  Potassium, change to high, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 10
  Potassium, change to high, Day 14 | 0 | 0 | 1 | 0
  Sodium, change to low, Day 7: number analyzed (Participants) | 14 | 15 | 12 | 13
  Sodium, change to low, Day 7 | 0 | 0 | 0 | 1
  Sodium, change to high, Day 7: number analyzed (Participants) | 14 | 15 | 12 | 13
  Sodium, change to high, Day 7 | 1 | 0 | 0 | 0
  Sodium, change to high, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 10
  Sodium, change to high, Day 14 | 1 | 0 | 0 | 0
  Total Bilirubin, change to high, Day 7: number analyzed (Participants) | 14 | 15 | 12 | 13
  Total Bilirubin, change to high, Day 7 | 0 | 0 | 0 | 1
  Total Protein, change to low, Day 7: number analyzed (Participants) | 14 | 15 | 12 | 13
  Total Protein, change to low, Day 7 | 1 | 0 | 1 | 0
  Total Protein, change to low, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 10
  Total Protein, change to low, Day 14 | 0 | 0 | 0 | 1
  Urea, change to high, Day 7: number analyzed (Participants) | 14 | 15 | 12 | 13
  Urea, change to high, Day 7 | 0 | 0 | 0 | 1
  Urea, change to low, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 10
  Urea, change to low, Day 14 | 0 | 1 | 0 | 1
  Uric acid, change to low, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 10
  Uric acid, change to low, Day 14 | 0 | 0 | 3 | 0
  Uric acid, change to high, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 10
  Uric acid, change to high, Day 14 | 0 | 1 | 0 | 0

17. Secondary Outcome: Number of Participants With Hematology Abnormal Change From Baseline Values Relative to the Normal Range at Day 7 and 14
Description: The parameters of biochemistry with their normal range included: basophils (0-0.2 giga cells [GI]/L), eosinophils (0.05-0.55 GI/L), haematocrit (0.41-0.5 ratio), hemoglobin (138-172 g/L), lymphocytes (0.85-4.1 GI/L), mean corpuscle hemoglobin ([MCH] 27-33 picogram [pg]), mean corpuscle hemoglobin concentration ([MCHC] 320-360 g/L), mean corpuscle volume ([MCV] 80-100 femtoliter [fl]), monocytes (0.2-1.1 GI/L), segmented neutrophils (1.8-8 GI/L), total neutrophils (1.8-8 GI/L), platelet count (130-400 GI/L), red blood cell ([RBC] 4.4-5.8 trillion cells [TI]/L) count and white blood cell ([WBC] 3.8-10.8 GI/L) count. The assessments were performed on Day 1, Day 7 and Day 14. Baseline was defined as the assessment done on Day 1. Only those parameters for which at least one value of abnormality (to low or to high) change from Baseline, relative to normal ranges were reported are summarized.
Time Frame: Baseline (Day 1) up to Day 14
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
Participants
  Eosinophils, change to low, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  Eosinophils, change to low, Day 7 | 0 | 0 | 1 | 0
  Eosinophils, change to high, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  Eosinophils, change to high, Day 7 | 0 | 1 | 0 | 1
  Eosinophils, change to high, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  Eosinophils, change to high, Day 14 | 0 | 0 | 1 | 1
  Hematocrit, change to low, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  Hematocrit, change to low, Day 7 | 0 | 0 | 1 | 0
  Hematocrit, change to high, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  Hematocrit, change to high, Day 7 | 0 | 0 | 0 | 1
  Hematocrit, change to low, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  Hematocrit, change to low, Day 14 | 1 | 0 | 1 | 0
  Hemoglobin, change to low, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  Hemoglobin, change to low, Day 7 | 0 | 0 | 2 | 0
  Hemoglobin, change to low, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  Hemoglobin, change to low, Day 14 | 0 | 0 | 2 | 0
  Lymphocytes, change to low, Day 7: number analyzed (Participants) | 14 | 14 | 13 | 13
  Lymphocytes, change to low, Day 7 | 1 | 0 | 0 | 0
  Lymphocytes, change to high, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  Lymphocytes, change to high, Day 7 | 1 | 0 | 0 | 0
  Lymphocytes, change to low, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  Lymphocytes, change to low, Day 14 | 1 | 0 | 0 | 0
  MCH, change to high, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  MCH, change to high, Day 7 | 0 | 0 | 1 | 1
  MCH, change to high, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  MCH, change to high, Day 14 | 0 | 1 | 0 | 0
  MCV, change to high, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  MCV, change to high, Day 7 | 0 | 0 | 0 | 1
  MCV, change to high, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  MCV, change to high, Day 14 | 0 | 0 | 1 | 0
  Monocytes, change to low, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  Monocytes, change to low, Day 7 | 1 | 0 | 1 | 1
  Monocytes, change to high, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  Monocytes, change to high, Day 7 | 0 | 0 | 0 | 1
  Monocytes, change to low, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  Monocytes, change to low, Day 14 | 0 | 0 | 0 | 1
  Monocytes, change to high, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  Monocytes, change to high, Day 14 | 0 | 0 | 0 | 1
  Platelet count, change to high, Day 14: number analyzed (Participants) | 13 | 15 | 12 | 9
  Platelet count, change to high, Day 14 | 1 | 0 | 0 | 0
  RBC count, change to low, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  RBC count, change to low, Day 7 | 0 | 1 | 1 | 0
  RBC count, change to low, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  RBC count, change to low, Day 14 | 0 | 1 | 1 | 0
  Segmented Neutrophils, change to low, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  Segmented Neutrophils, change to low, Day 7 | 1 | 0 | 0 | 0
  Segmented Neutrophils, change to high, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  Segmented Neutrophils, change to high, Day 7 | 1 | 1 | 0 | 0
  Segmented Neutrophils, change to low, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  Segmented Neutrophils, change to low, Day 14 | 0 | 0 | 1 | 1
  Segmented Neutrophils, change to high, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  Segmented Neutrophils, change to high, Day 14 | 1 | 0 | 1 | 0
  Total Neutrophils, change to low, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  Total Neutrophils, change to low, Day 7 | 1 | 0 | 0 | 0
  Total Neutrophils, change to high, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  Total Neutrophils, change to high, Day 7 | 1 | 1 | 0 | 0
  Total Neutrophils, change to low, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  Total Neutrophils, change to low, Day 14 | 0 | 0 | 1 | 1
  Total Neutrophils, change to high, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  Total Neutrophils, change to high, Day 14 | 1 | 0 | 1 | 0
  WBC count, change to low, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  WBC count, change to low, Day 7 | 2 | 0 | 0 | 0
  WBC count, change to high, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  WBC count, change to high, Day 7 | 0 | 0 | 0 | 1
  WBC count, change to low, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  WBC count, change to low, Day 14 | 1 | 0 | 0 | 0
  WBC count, change to high, Day 14: number analyzed (Participants) | 14 | 15 | 12 | 10
  WBC count, change to high, Day 14 | 1 | 0 | 1 | 0

18. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) at Pre-dose, Weighted Mean FEV1 at 0-4 h and Maximum FEV1 0-4 h Over Time
Description: FEV1 is defined as the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEV1 was assessed pre-dose at Day 1, 2, 7, 8, 14 and 15. FEV1 was assessed post-dose at Day 1, 2, 7, 8 and 14. Lung function test of FEV1 was performed at the approximately same time at each visit in the morning and highest of the 3 measurements were recorded. Baseline was defined as the assessment done on pre-dose Day 1. The change from Baseline pre-dose was calculated by subtracting the Baseline value (pre-dose Day 1) from the individual post Baseline (Day 2, 7, 8, 14 and 15) values. Weighted mean was calculated by calculating the AUC, and then dividing by the relevant time interval. AUC was calculated using the trapezoidal rule. The weighted mean FEV1 0-4 h change from Baseline was the AAUCMB obtained at Day 1, 2, 7, 8, 14 and 15. The maximum FEV1 0-4 h change from Baseline was obtained at Day 1, Day 2, Day 7, Day 8, Day 14 and Day 15.
Time Frame: Baseline (Day 1, pre-dose) up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Litres (L)
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
Litres (L)
  Day 7, Pre-dose: number analyzed (Participants) | 15 | 15 | 13 | 14
  Day 7, Pre-dose | -0.019 (0.3068) | 0.139 (0.1159) | 0.149 (0.1934) | 0.181 (0.2584)
  Day 14, Pre-dose: number analyzed (Participants) | 14 | 15 | 12 | 12
  Day 14, Pre-dose | -0.006 (0.2975) | 0.155 (0.1449) | 0.183 (0.2502) | 0.055 (0.2349)
  Weighted mean 0-4 h, Day 1: number analyzed (Participants) | 15 | 15 | 16 | 16
  Weighted mean 0-4 h, Day 1 | 0.0513 (0.11220) | 0.1794 (0.10171) | 0.2099 (0.14168) | 0.2012 (0.12209)
  Weighted mean 0-4 h, Day 2: number analyzed (Participants) | 15 | 16 | 16 | 16
  Weighted mean 0-4 h, Day 2 | 0.0609 (0.17522) | 0.2427 (0.11735) | 0.2890 (0.17558) | 0.1829 (0.26427)
  Weighted mean 0-4 h, Day 7: number analyzed (Participants) | 15 | 15 | 13 | 14
  Weighted mean 0-4 h, Day 7 | 0.0480 (0.24623) | 0.2001 (0.12189) | 0.2463 (0.19308) | 0.2195 (0.23573)
  Weighted mean 0-4 h, Day 8: number analyzed (Participants) | 15 | 14 | 13 | 13
  Weighted mean 0-4 h, Day 8 | 0.0563 (0.25677) | 0.2313 (0.12148) | 0.2419 (0.17906) | 0.1542 (0.26356)
  Weighted mean 0-4 h, Day 14: number analyzed (Participants) | 13 | 15 | 12 | 12
  Weighted mean 0-4 h, Day 14 | 0.0557 (0.27371) | 0.1899 (0.13425) | 0.2798 (0.25865) | 0.1290 (0.29444)
  Weighted mean 0-4 h, Day 15: number analyzed (Participants) | 15 | 13 | 12 | 13
  Weighted mean 0-4 h, Day 15 | 0.0339 (0.25474) | 0.2096 (0.10678) | 0.1973 (0.16988) | 0.1938 (0.28321)
  Maximum 0-4 h, Day 1: number analyzed (Participants) | 16 | 16 | 16 | 17
  Maximum 0-4 h, Day 1 | 0.125 (0.1348) | 0.241 (0.1191) | 0.276 (0.1587) | 0.272 (0.1500)
  Maximum 0-4 h, Day 2: number analyzed (Participants) | 15 | 16 | 16 | 16
  Maximum 0-4 h, Day 2 | 0.152 (0.1888) | 0.285 (0.1254) | 0.356 (0.1853) | 0.264 (0.2887)
  Maximum 0-4 h, Day 7: number analyzed (Participants) | 15 | 15 | 13 | 14
  Maximum 0-4 h, Day 7 | 0.137 (0.2752) | 0.251 (0.1196) | 0.317 (0.2080) | 0.283 (0.2459)
  Maximum 0-4 h, Day 8: number analyzed (Participants) | 15 | 15 | 13 | 13
  Maximum 0-4 h, Day 8 | 0.133 (0.2888) | 0.277 (0.1150) | 0.295 (0.1852) | 0.224 (0.2524)
  Maximum 0-4 h, Day 14: number analyzed (Participants) | 15 | 15 | 12 | 13
  Maximum 0-4 h, Day 14 | 0.093 (0.2785) | 0.227 (0.1391) | 0.332 (0.2697) | 0.191 (0.2881)
  Maximum 0-4 h, Day 15: number analyzed (Participants) | 15 | 15 | 12 | 13
  Maximum 0-4 h, Day 15 | 0.121 (0.2500) | 0.245 (0.1445) | 0.289 (0.1721) | 0.283 (0.2909)

19. Secondary Outcome: Mean FEV1 Weighted Mean FEV1 at 0-4 h and Maximum FEV1 at 0-4 h Over Time
Description: FEV1 is defined as the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEV1 was assessed pre-dose and post-dose at Day 1, 2, 7, 8, 14 and 15. Lung function test of FEV1 was performed at the approximately same time at each visit in the morning and highest of the 3 measurements were recorded. Weighted mean was calculated by calculating the AUC, and then dividing by the relevant time interval. AUC was calculated using the trapezoidal rule. The weighted mean FEV1 0-4 h and maximum FEV1 0-4 h was obtained at Day 1, 2, 7, 8, 14 and 15.
Time Frame: Day 1 up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
L
  Weighted mean 0-4, Day 1: number analyzed (Participants) | 15 | 15 | 16 | 16
  Weighted mean 0-4, Day 1 | 1.6180 (0.49986) | 1.5294 (0.49878) | 2.0224 (0.62567) | 1.6674 (0.47398)
  Weighted mean 0-4, Day 2: number analyzed (Participants) | 16 | 16 | 16 | 17
  Weighted mean 0-4, Day 2 | 1.6498 (0.44952) | 1.5796 (0.52525) | 2.1015 (0.62389) | 1.6480 (0.53142)
  Weighted mean 0-4, Day 7: number analyzed (Participants) | 16 | 15 | 14 | 15
  Weighted mean 0-4, Day 7 | 1.6261 (0.43336) | 1.5427 (0.51959) | 2.0355 (0.61827) | 1.7053 (0.52221)
  Weighted mean 0-4, Day 8: number analyzed (Participants) | 16 | 14 | 14 | 14
  Weighted mean 0-4, Day 8 | 1.6375 (0.53044) | 1.6027 (0.51660) | 2.0637 (0.61246) | 1.6599 (0.51218)
  Weighted mean 0-4, Day 14: number analyzed (Participants) | 14 | 15 | 13 | 12
  Weighted mean 0-4, Day 14 | 1.6861 (0.50464) | 1.5326 (0.51142) | 2.1411 (0.61845) | 1.6457 (0.61933)
  Weighted mean 0-4, Day 15: number analyzed (Participants) | 16 | 13 | 13 | 14
  Weighted mean 0-4, Day 15 | 1.6155 (0.49847) | 1.4719 (0.47004) | 2.0638 (0.53939) | 1.6611 (0.51360)
  Maximum 0-4 h, Day 1: number analyzed (Participants) | 17 | 16 | 16 | 18
  Maximum 0-4 h, Day 1 | 1.698 (0.4811) | 1.578 (0.5034) | 2.089 (0.6341) | 1.708 (0.4848)
  Maximum 0-4 h, Day 2: number analyzed (Participants) | 16 | 16 | 16 | 17
  Maximum 0-4 h, Day 2 | 1.741 (0.4597) | 1.622 (0.5329) | 2.168 (0.6217) | 1.726 (0.5514)
  Maximum 0-4 h, Day 7: number analyzed (Participants) | 16 | 15 | 14 | 15
  Maximum 0-4 h, Day 7 | 1.712 (0.4639) | 1.593 (0.5196) | 2.104 (0.6429) | 1.766 (0.5245)
  Maximum 0-4 h, Day 8: number analyzed (Participants) | 16 | 15 | 14 | 14
  Maximum 0-4 h, Day 8 | 1.717 (0.5510) | 1.620 (0.5182) | 2.120 (0.6170) | 1.729 (0.5083)
  Maximum 0-4 h, Day 14: number analyzed (Participants) | 16 | 15 | 13 | 14
  Maximum 0-4 h, Day 14 | 1.684 (0.5236) | 1.569 (0.5193) | 2.203 (0.6287) | 1.664 (0.5901)
  Maximum 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 13 | 14
  Maximum 0-4 h, Day 15 | 1.704 (0.5020) | 1.587 (0.5060) | 2.156 (0.5717) | 1.745 (0.5673)

20. Secondary Outcome: Change From Baseline in Weighted Mean FEV1 Over 22- 24 h on Days 1, 7 and 14
Description: FEV1 is defined as the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Lung function test of FEV1 was performed at the approximately same time at each visit in the morning and highest of the 3 measurements were recorded. Weighted mean was calculated by calculating the AUC, and then dividing by the relevant time interval. AUC was calculated using the trapezoidal rule. The weighted mean FEV1 over 22-24 h was obtained at Day 1, Day 7 and Day 14 which was recorded up to Day 2, Day 8 and Day 15. Baseline was defined as the assessment on Day 1 pre-dose. Change from Baseline was calculated by subtracting the Baseline (Day 1, pre-dose) value from the individual post Baseline (Day 1, Day 7 and Day 14) values.
Time Frame: Baseline (Day 1, pre-dose) up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
L
  Day 1: number analyzed (Participants) | 15 | 16 | 16 | 16
  Day 1 | 0.0191 (0.04224) | 0.1322 (0.04171) | 0.1781 (0.04194) | 0.0955 (0.04043)
  Day 7: number analyzed (Participants) | 15 | 14 | 13 | 13
  Day 7 | -0.0174 (0.05640) | 0.1568 (0.05818) | 0.1539 (0.06073) | 0.1204 (0.05723)
  Day 14: number analyzed (Participants) | 15 | 13 | 12 | 13
  Day 14 | -0.0225 (0.05719) | 0.1166 (0.06178) | 0.1681 (0.06615) | 0.0732 (0.05827)
Statistical Analysis 1: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for FEV1 over 22-24 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline FEV1, gender, age and treatment; Mean Difference (Net) = 0.1131, 95% CI 2-sided [-0.0031 to 0.2293]
Statistical Analysis 2: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for FEV1 over 22-24 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline FEV1, gender, age and treatment; Mean Difference (Net) = 0.1590, 95% CI 2-sided [0.0408 to 0.2771]
Statistical Analysis 3: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for FEV1 over 22-24 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline FEV1, gender, age and treatment; Mean Difference (Net) = 0.0764, 95% CI 2-sided [-0.0375 to 0.1903]
Statistical Analysis 4: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for FEV1 over 22-24 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline FEV1, gender, age and treatment; Mean Difference (Net) = 0.1741, 95% CI 2-sided [0.0178 to 0.3305]
Statistical Analysis 5: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for FEV1 over 22-24 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline FEV1, gender, age and treatment; Mean Difference (Net) = 0.1713, 95% CI 2-sided [0.0060 to 0.3365]
Statistical Analysis 6: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for FEV1 over 22-24 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline FEV1, gender, age and treatment; Mean Difference (Net) = 0.1377, 95% CI 2-sided [-0.0233 to 0.2987]
Statistical Analysis 7: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for FEV1 over 22-24 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline FEV1, gender, age and treatment; Mean Difference (Net) = 0.1390, 95% CI 2-sided [-0.0266 to 0.3046]
Statistical Analysis 8: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for FEV1 over 22-24 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline FEV1, gender, age and treatment; Mean Difference (Net) = 0.1906, 95% CI 2-sided [0.0177 to 0.3635]
Statistical Analysis 9: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for FEV1 over 22-24 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline FEV1, gender, age and treatment; Mean Difference (Net) = 0.0956, 95% CI 2-sided [-0.0686 to 0.2599]

21. Secondary Outcome: Mean Morning and Evening Peak Expiratory Flow Rate (PEFR) Over Time
Description: PEF is a measure of lung function and measures how fast a person can breathe out. It was measured using a peak flow meter by the participants and recorded on daily record cards each day in the morning and evening from Screening up to Follow-up. The morning measurements were performed prior to the participant taking the morning dose of study medication or rescue medication. The evening measurements were performed prior to the participant taking the evening dose of study medication or rescue medication. The highest of the 3 values of morning and evening PEF were recorded on the diary card. The mean of 7 days of each morning and evening measurements were reported for the Run-in Week, Week 1, Week 2 and Follow-up.
Time Frame: Up to Follow-up (Day 17)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Liters per minute (L/min)
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
Liters per minute (L/min)
  Morning PEFR, Run-in: number analyzed (Participants) | 17 | 15 | 17 | 18
  Morning PEFR, Run-in | 268.20 (85.986) | 249.99 (78.848) | 276.45 (95.245) | 244.44 (52.722)
  Morning PEFR, Week 1: number analyzed (Participants) | 16 | 16 | 17 | 17
  Morning PEFR, Week 1 | 271.37 (85.186) | 266.22 (61.112) | 299.22 (99.017) | 254.39 (63.273)
  Morning PEFR, Week 2: number analyzed (Participants) | 16 | 15 | 14 | 14
  Morning PEFR, Week 2 | 264.52 (89.793) | 265.23 (66.178) | 295.75 (106.748) | 257.84 (74.086)
  Morning PEFR, Follow-up: number analyzed (Participants) | 16 | 15 | 13 | 14
  Morning PEFR, Follow-up | 270.16 (95.536) | 262.83 (55.709) | 297.69 (111.329) | 264.64 (83.106)
  Evening PEFR, Run-in: number analyzed (Participants) | 17 | 15 | 16 | 18
  Evening PEFR, Run-in | 266.76 (79.352) | 251.85 (63.927) | 270.10 (93.699) | 252.64 (66.592)
  Evening PEFR, Week 1: number analyzed (Participants) | 16 | 16 | 17 | 17
  Evening PEFR, Week 1 | 273.45 (82.356) | 278.80 (65.325) | 311.46 (99.984) | 264.45 (78.755)
  Evening PEFR, Week 2: number analyzed (Participants) | 16 | 15 | 14 | 14
  Evening PEFR, Week 2 | 274.13 (84.622) | 275.12 (59.122) | 302.04 (110.097) | 263.01 (88.672)
  Evening PEFR, Follow-up: number analyzed (Participants) | 12 | 14 | 11 | 9
  Evening PEFR, Follow-up | 284.75 (84.680) | 262.14 (55.737) | 319.09 (110.336) | 314.44 (99.858)

22. Secondary Outcome: Mean Use of Rescue Medication Over Period
Description: Ipratropium bromide was provided as the rescue medication. The use of rescue medication was recorded by the participants on daily record cards each day in the morning and evening from Screening up to Follow-up. The mean of 7 days (puffs per 24 h) were reported for the Run-in Week, Week 1, Week 2 and Follow-up.
Time Frame: Up to Follow-up (Day 17)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Puffs per 24 h
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
Puffs per 24 h
  Run-in: number analyzed (Participants) | 15 | 14 | 10 | 16
  Run-in | 3.12 (2.525) | 2.46 (2.464) | 1.38 (1.554) | 1.66 (1.363)
  Week 1: number analyzed (Participants) | 16 | 12 | 13 | 12
  Week 1 | 1.99 (2.453) | 1.63 (1.755) | 0.73 (1.133) | 1.25 (2.003)
  Week 2: number analyzed (Participants) | 16 | 11 | 12 | 10
  Week 2 | 2.24 (3.053) | 1.61 (2.021) | 0.79 (1.159) | 0.93 (0.962)
  Follow-up: number analyzed (Participants) | 12 | 13 | 9 | 7
  Follow-up | 2.17 (2.552) | 1.38 (1.502) | 1.11 (1.364) | 0.86 (1.574)

23. Secondary Outcome: Number of Participants With Rescue Free Days
Description: Ipratropium bromide was provided as the rescue medication. The use of rescue medication was recorded by the participants on daily record cards each day in the morning and evening from Screening up to Follow-up. The percentage of rescue free days during the Run-in week, Week 1, Week 2 and Follow-up Week were assessed. Data is reported for number of participants with < 20%, >=20 to <40%, >=40 to <60%, >=60 to <80% and >=80% rescue free days.
Time Frame: Up to Follow-up (Day 17)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
Participants
  Run-in: number analyzed (Participants) | 15 | 14 | 10 | 16
  Run-in: < 20% | 10 | 9 | 5 | 10
  Run-in: >=20 to <40% | 0 | 2 | 1 | 0
  Run-in: >=40 to <60% | 3 | 0 | 0 | 2
  Run-in: >=60 to <80% | 1 | 0 | 0 | 1
  Run-in: >=80% | 1 | 3 | 4 | 3
  Week 1: number analyzed (Participants) | 16 | 12 | 13 | 12
  Week 1: < 20% | 7 | 5 | 3 | 4
  Week 1: >=20 to <40% | 1 | 1 | 0 | 0
  Week 1: >=40 to <60% | 2 | 1 | 3 | 1
  Week 1: >=60 to <80% | 0 | 0 | 1 | 1
  Week 1: >=80% | 6 | 5 | 6 | 6
  Week 2: number analyzed (Participants) | 16 | 11 | 12 | 10
  Week 2: < 20% | 7 | 4 | 3 | 3
  Week 2: >=20 to <40% | 1 | 1 | 1 | 0
  Week 2: >=40 to <60% | 1 | 0 | 1 | 2
  Week 2: >=60 to <80% | 1 | 1 | 2 | 2
  Week 2: >=80% | 6 | 5 | 5 | 3
  Follow-up: number analyzed (Participants) | 12 | 13 | 9 | 7
  Follow-up: < 20% | 9 | 8 | 5 | 2
  Follow-up: >=20 to <40% | 0 | 0 | 0 | 0
  Follow-up: >=40 to <60% | 0 | 0 | 0 | 0
  Follow-up: >=60 to <80% | 0 | 0 | 0 | 0
  Follow-up: >=80% | 3 | 5 | 4 | 5

24. Secondary Outcome: Change From Baseline in Pre-dose Fasting Glucose and Potassium at Day 7 and 14
Description: Blood samples were collected at pre-dose on Day 1, Day 7 and Day 14. Baseline was defined as the assessment done on pre-dose, Day 1. Change from Baseline was calculated by subtracting the Baseline (Day 1, pre-dose) value from the individual post Baseline (Day 7 and Day 14) values.
Time Frame: Baseline (Day 1, pre-dose) up to Day 14
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimole (mmol)/L)
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
Millimole (mmol)/L)
  Fasting Glucose, Day 7: number analyzed (Participants) | 16 | 15 | 12 | 15
  Fasting Glucose, Day 7 | -0.22 (0.742) | 0.61 (1.175) | 0.11 (0.673) | 0.22 (1.103)
  Fasting Glucose, Day 14: number analyzed (Participants) | 15 | 15 | 13 | 14
  Fasting Glucose, Day 14 | 0.08 (1.229) | 0.57 (0.856) | 0.19 (0.639) | 0.13 (1.040)
  Fasting Potassium, Day 7: number analyzed (Participants) | 15 | 12 | 10 | 12
  Fasting Potassium, Day 7 | 0.22 (0.328) | -0.11 (0.436) | 0.03 (0.675) | 0.17 (0.737)
  Fasting Potassium, Day 14: number analyzed (Participants) | 15 | 12 | 12 | 11
  Fasting Potassium, Day 14 | 0.00 (0.285) | -0.16 (0.500) | 0.02 (0.354) | 0.33 (0.504)

25. Secondary Outcome: Change From Baseline in Weighted Mean Glucose and Potassium 0-4 h, Maximum Glucose 0-4 h and Minimum Potassium 0-4 h Over Time
Description: Blood samples were collected at pre-dose and 4 h post-dose on Day 1, Day 2, Day 7, Day 8, Day 14 and Day 15. Weighted mean was calculated by calculating the AUC, and then dividing by the relevant time interval. AUC was calculated using the trapezoidal rule. Baseline was defined as the assessment on Day 1 pre-dose. The weighted mean change from Baseline was the AAUCMB. Change from Baseline in maximum glucose 0-4 h and minimum potassium 0-4 h was calculated by subtracting the Baseline (Day 1, pre-dose) value from the individual post Baseline (Day 1 to Day 15) values.
Time Frame: Baseline (Day 1, pre-dose) up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
mmol/L
  Weighted Mean Glucose 0-4 h, Day 1: number analyzed (Participants) | 16 | 16 | 16 | 17
  Weighted Mean Glucose 0-4 h, Day 1 | 0.048 (0.2097) | 0.057 (0.2061) | 0.285 (0.2068) | 0.140 (0.1946)
  Weighted Mean Glucose 0-4 h, Day 2: number analyzed (Participants) | 15 | 15 | 15 | 16
  Weighted Mean Glucose 0-4 h, Day 2 | -0.137 (0.2749) | 0.062 (0.2689) | 0.497 (0.2711) | -0.072 (0.2550)
  Weighted Mean Glucose 0-4 h, Day 7: number analyzed (Participants) | 16 | 15 | 11 | 15
  Weighted Mean Glucose 0-4 h, Day 7 | -0.002 (0.1978) | 0.095 (0.1994) | 0.406 (0.2349) | 0.078 (0.1929)
  Weighted Mean Glucose 0-4 h, Day 8: number analyzed (Participants) | 16 | 14 | 11 | 14
  Weighted Mean Glucose 0-4 h, Day 8 | -0.183 (0.3111) | 0.061 (0.3200) | 0.613 (0.3614) | -0.039 (0.3097)
  Weighted Mean Glucose 0-4 h, Day 14: number analyzed (Participants) | 15 | 14 | 11 | 14
  Weighted Mean Glucose 0-4 h, Day 14 | 0.193 (0.2104) | 0.250 (0.2046) | 0.055 (0.2309) | 0.006 (0.1956)
  Weighted Mean Glucose 0-4 h, Day 15: number analyzed (Participants) | 15 | 15 | 12 | 14
  Weighted Mean Glucose 0-4 h, Day 15 | -0.100 (0.2505) | -0.006 (0.2404) | 0.258 (0.2737) | 0.078 (0.2413)
  Weighted Mean Potassium 0-4 h, Day 1: number analyzed (Participants) | 16 | 13 | 15 | 13
  Weighted Mean Potassium 0-4 h, Day 1 | 0.183 (0.0999) | -0.110 (0.1062) | -0.188 (0.1016) | 0.030 (0.1063)
  Weighted Mean Potassium 0-4 h, Day 2: number analyzed (Participants) | 14 | 12 | 13 | 13
  Weighted Mean Potassium 0-4 h, Day 2 | 0.376 (0.1575) | 0.160 (0.1634) | -0.160 (0.1609) | 0.358 (0.1576)
  Weighted Mean Potassium 0-4 h, Day 7: number analyzed (Participants) | 15 | 12 | 9 | 12
  Weighted Mean Potassium 0-4 h, Day 7 | 0.267 (0.1318) | -0.219 (0.1421) | -0.295 (0.1664) | 0.077 (0.1415)
  Weighted Mean Potassium 0-4 h, Day 8: number analyzed (Participants) | 15 | 12 | 9 | 11
  Weighted Mean Potassium 0-4 h, Day 8 | 0.247 (0.1051) | 0.322 (0.1115) | -0.027 (0.1311) | 0.350 (0.1154)
  Weighted Mean Potassium 0-4 h, Day 14: number analyzed (Participants) | 15 | 11 | 10 | 11
  Weighted Mean Potassium 0-4 h, Day 14 | 0.218 (0.1140) | -0.081 (0.1233) | -0.053 (0.1325) | 0.123 (0.1224)
  Weighted Mean Potassium 0-4 h, Day 15: number analyzed (Participants) | 15 | 12 | 11 | 11
  Weighted Mean Potassium 0-4 h, Day 15 | 0.155 (0.1120) | 0.328 (0.1197) | -0.041 (0.1276) | 0.293 (0.1234)
  Maximum Glucose 0-4 h, Day 1 | 0.65 (0.361) | 0.51 (0.365) | 0.94 (0.357) | 0.48 (0.336)
  Maximum Glucose 0-4 h, Day 2: number analyzed (Participants) | 16 | 16 | 17 | 17
  Maximum Glucose 0-4 h, Day 2 | 0.21 (0.363) | 0.61 (0.357) | 0.89 (0.350) | 0.44 (0.337)
  Maximum Glucose 0-4 h, Day 7: number analyzed (Participants) | 16 | 15 | 13 | 15
  Maximum Glucose 0-4 h, Day 7 | 0.52 (0.367) | 0.47 (0.368) | 1.05 (0.402) | 0.65 (0.359)
  Maximum Glucose 0-4 h, Day 8: number analyzed (Participants) | 16 | 15 | 13 | 14
  Maximum Glucose 0-4 h, Day 8 | 0.28 (0.431) | 0.53 (0.425) | 1.13 (0.464) | 0.60 (0.429)
  Maximum Glucose 0-4 h, Day 14: number analyzed (Participants) | 16 | 15 | 13 | 14
  Maximum Glucose 0-4 h, Day 14 | 0.37 (0.434) | 0.42 (0.431) | 1.12 (0.473) | 0.37 (0.433)
  Maximum Glucose 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 12 | 14
  Maximum Glucose 0-4 h, Day 15 | 0.21 (0.348) | 0.43 (0.345) | 1.05 (0.392) | 0.70 (0.346)
  Minimum Potassium 0-4 h, Day 1: number analyzed (Participants) | 17 | 13 | 16 | 15
  Minimum Potassium 0-4 h, Day 1 | -0.12 (0.094) | -0.31 (0.104) | -0.35 (0.095) | -0.32 (0.096)
  Minimum Potassium 0-4 h, Day 2: number analyzed (Participants) | 16 | 13 | 16 | 14
  Minimum Potassium 0-4 h, Day 2 | 0.07 (0.127) | -0.03 (0.135) | -0.31 (0.125) | 0.05 (0.130)
  Minimum Potassium 0-4 h, Day 7: number analyzed (Participants) | 16 | 12 | 12 | 12
  Minimum Potassium 0-4 h, Day 7 | 0.07 (0.143) | -0.47 (0.158) | -0.47 (0.161) | -0.27 (0.156)
  Minimum Potassium 0-4 h, Day 8: number analyzed (Participants) | 16 | 12 | 12 | 11
  Minimum Potassium 0-4 h, Day 8 | 0.09 (0.099) | 0.13 (0.109) | -0.30 (0.111) | 0.13 (0.113)
  Minimum Potassium 0-4 h, Day 14: number analyzed (Participants) | 16 | 12 | 12 | 11
  Minimum Potassium 0-4 h, Day 14 | -0.06 (0.091) | -0.21 (0.100) | -0.29 (0.103) | -0.12 (0.103)
  Minimum Potassium 0-4 h, Day 15: number analyzed (Participants) | 16 | 12 | 11 | 11
  Minimum Potassium 0-4 h, Day 15 | -0.02 (0.099) | 0.03 (0.109) | -0.37 (0.117) | 0.02 (0.113)
Statistical Analysis 1: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for weighted mean glucose 0-4 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.009, 95% CI 2-sided [-0.590 to 0.608]
Statistical Analysis 2: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for weighted mean glucose 0-4 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.237, 95% CI 2-sided [-0.354 to 0.829]
Statistical Analysis 3: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for weighted mean glucose 0-4 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.093, 95% CI 2-sided [-0.469 to 0.654]
Statistical Analysis 4: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for weighted mean glucose 0-4 h at Day 2; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.199, 95% CI 2-sided [-0.591 to 0.988]
Statistical Analysis 5: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for weighted mean glucose 0-4 h at Day 2; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.633, 95% CI 2-sided [-0.152 to 1.418]
Statistical Analysis 6: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for weighted mean glucose 0-4 h at Day 2; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.065, 95% CI 2-sided [-0.667 to 0.797]
Statistical Analysis 7: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for weighted mean glucose 0-4 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.097, 95% CI 2-sided [-0.476 to 0.670]
Statistical Analysis 8: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for weighted mean glucose 0-4 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.408, 95% CI 2-sided [-0.208 to 1.024]
Statistical Analysis 9: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for weighted mean glucose 0-4 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.080, 95% CI 2-sided [-0.471 to 0.631]
Statistical Analysis 10: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for weighted mean glucose 0-4 h at Day 8; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.245, 95% CI 2-sided [-0.660 to 1.149]
Statistical Analysis 11: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for weighted mean glucose 0-4 h at Day 8; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.796, 95% CI 2-sided [-0.174 to 1.766]
Statistical Analysis 12: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for weighted mean glucose 0-4 h at Day 8; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.144, 95% CI 2-sided [-0.742 to 1.030]
Statistical Analysis 13: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for weighted mean glucose 0-4 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.056, 95% CI 2-sided [-0.556 to 0.669]
Statistical Analysis 14: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for weighted mean glucose 0-4 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = -0.138, 95% CI 2-sided [-0.767 to 0.491]
Statistical Analysis 15: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for weighted mean glucose 0-4 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = -0.187, 95% CI 2-sided [-0.765 to 0.391]
Statistical Analysis 16: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for weighted mean glucose 0-4 h at Day 15; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.094, 95% CI 2-sided [-0.619 to 0.806]
Statistical Analysis 17: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for weighted mean glucose 0-4 h at Day 15; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.358, 95% CI 2-sided [-0.390 to 1.105]
Statistical Analysis 18: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for weighted mean glucose 0-4 h at Day 15; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.178, 95% CI 2-sided [-0.522 to 0.877]
Statistical Analysis 19: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for weighted mean potassium 0-4 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.294, 95% CI 2-sided [-0.586 to -0.001]
Statistical Analysis 20: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for weighted mean potassium 0-4 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.371, 95% CI 2-sided [-0.657 to -0.085]
Statistical Analysis 21: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for weighted mean potassium 0-4 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.153, 95% CI 2-sided [-0.440 to 0.133]
Statistical Analysis 22: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for weighted mean potassium 0-4 h at Day 2; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.216, 95% CI 2-sided [-0.679 to 0.247]
Statistical Analysis 23: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for weighted mean potassium 0-4 h at Day 2; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.536, 95% CI 2-sided [-0.998 to -0.074]
Statistical Analysis 24: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for weighted mean potassium 0-4 h at Day 2; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.018, 95% CI 2-sided [-0.452 to 0.416]
Statistical Analysis 25: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for weighted mean potassium 0-4 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.486, 95% CI 2-sided [-0.878 to -0.095]
Statistical Analysis 26: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for weighted mean potassium 0-4 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.562, 95% CI 2-sided [-0.990 to -0.135]
Statistical Analysis 27: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for weighted mean potassium 0-4 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.190, 95% CI 2-sided [-0.575 to 0.196]
Statistical Analysis 28: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for weighted mean potassium 0-4 h at Day 8; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = 0.075, 95% CI 2-sided [-0.235 to 0.385]
Statistical Analysis 29: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for weighted mean potassium 0-4 h at Day 8; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.275, 95% CI 2-sided [-0.623 to 0.073]
Statistical Analysis 30: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for weighted mean potassium 0-4 h at Day 8; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = 0.103, 95% CI 2-sided [-0.213 to 0.418]
Statistical Analysis 31: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for weighted mean potassium 0-4 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.299, 95% CI 2-sided [-0.640 to 0.042]
Statistical Analysis 32: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for weighted mean potassium 0-4 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.271, 95% CI 2-sided [-0.621 to 0.079]
Statistical Analysis 33: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for weighted mean potassium 0-4 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.095, 95% CI 2-sided [-0.432 to 0.243]
Statistical Analysis 34: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for weighted mean potassium 0-4 h at Day 15; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = 0.173, 95% CI 2-sided [-0.158 to 0.505]
Statistical Analysis 35: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for weighted mean potassium 0-4 h at Day 15; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.196, 95% CI 2-sided [-0.535 to 0.143]
Statistical Analysis 36: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for weighted mean potassium 0-4 h at Day 15; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = 0.139, 95% CI 2-sided [-0.198 to 0.475]
Statistical Analysis 37: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for maximum glucose 0-4 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = -0.14, 95% CI 2-sided [-1.18 to 0.90]
Statistical Analysis 38: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for maximum glucose 0-4 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.29, 95% CI 2-sided [-0.72 to 1.30]
Statistical Analysis 39: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for maximum glucose 0-4 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = -0.17, 95% CI 2-sided [-1.15 to 0.80]
Statistical Analysis 40: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for maximum glucose 0-4 h at Day 2; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.40, 95% CI 2-sided [-0.64 to 1.44]
Statistical Analysis 41: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for maximum glucose 0-4 h at Day 2; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.69, 95% CI 2-sided [-0.32 to 1.70]
Statistical Analysis 42: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for maximum glucose 0-4 h at Day 2; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.23, 95% CI 2-sided [-0.74 to 1.20]
Statistical Analysis 43: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for maximum glucose 0-4 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = -0.05, 95% CI 2-sided [-1.11 to 1.01]
Statistical Analysis 44: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for maximum glucose 0-4 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.53, 95% CI 2-sided [-0.57 to 1.62]
Statistical Analysis 45: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for maximum glucose 0-4 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.89 to 1.15]
Statistical Analysis 46: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for maximum glucose 0-4 h at Day 8; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.26, 95% CI 2-sided [-0.98 to 1.50]
Statistical Analysis 47: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for maximum glucose 0-4 h at Day 8; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.86, 95% CI 2-sided [-0.42 to 2.14]
Statistical Analysis 48: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for maximum glucose 0-4 h at Day 8; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.32, 95% CI 2-sided [-0.90 to 1.54]
Statistical Analysis 49: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for maximum glucose 0-4 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.05, 95% CI 2-sided [-1.20 to 1.30]
Statistical Analysis 50: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for maximum glucose 0-4 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.75, 95% CI 2-sided [-0.53 to 2.03]
Statistical Analysis 51: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for maximum glucose 0-4 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.00, 95% CI 2-sided [-1.23 to 1.23]
Statistical Analysis 52: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for maximum glucose 0-4 h at Day 15; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.22, 95% CI 2-sided [-0.78 to 1.23]
Statistical Analysis 53: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for maximum glucose 0-4 h at Day 15; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.84, 95% CI 2-sided [-0.21 to 1.89]
Statistical Analysis 54: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for maximum glucose 0-4 h at Day 15; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline glucose, gender, age and treatment; Mean Difference (Net) = 0.49, 95% CI 2-sided [-0.50 to 1.48]
Statistical Analysis 55: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for minimum potassium 0-4 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.47 to 0.09]
Statistical Analysis 56: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for minimum potassium 0-4 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.49 to 0.04]
Statistical Analysis 57: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for minimum potassium 0-4 h at Day 1; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.46 to 0.07]
Statistical Analysis 58: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for minimum potassium 0-4 h at Day 2; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.47 to 0.27]
Statistical Analysis 59: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for minimum potassium 0-4 h at Day 2; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.38, 95% CI 2-sided [-0.73 to -0.03]
Statistical Analysis 60: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for minimum potassium 0-4 h at Day 2; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.37 to 0.34]
Statistical Analysis 61: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for minimum potassium 0-4 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.54, 95% CI 2-sided [-0.97 to -0.12]
Statistical Analysis 62: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for minimum potassium 0-4 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.55, 95% CI 2-sided [-0.98 to -0.12]
Statistical Analysis 63: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for minimum potassium 0-4 h at Day 7; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.34, 95% CI 2-sided [-0.76 to 0.08]
Statistical Analysis 64: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for minimum potassium 0-4 h at Day 8; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.26 to 0.33]
Statistical Analysis 65: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for minimum potassium 0-4 h at Day 8; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.40, 95% CI 2-sided [-0.70 to -0.10]
Statistical Analysis 66: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for minimum potassium 0-4 h at Day 8; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.26 to 0.34]
Statistical Analysis 67: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for minimum potassium 0-4 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.42 to 0.12]
Statistical Analysis 68: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for minimum potassium 0-4 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.51 to 0.04]
Statistical Analysis 69: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for minimum potassium 0-4 h at Day 14; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.34 to 0.21]
Statistical Analysis 70: Comparison: Placebo vs GW642444 100 mcg Once Daily; Placebo versus GW642444 100 mcg once daily for minimum potassium 0-4 h at Day 15; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.25 to 0.35]
Statistical Analysis 71: Comparison: Placebo vs GW642444 400 mcg Once Daily; Placebo versus GW642444 400 mcg once daily for minimum potassium 0-4 h at Day 15; Test type: Superiority; Regression, Linear; Mean Difference (Net) = -0.35, 95% CI 2-sided [-0.66 to -0.05]
Statistical Analysis 72: Comparison: Placebo vs Salmeterol 50 mcg BD; Placebo versus Salmeterol 50 mcg BD for minimum potassium 0-4 h at Day 15; Test type: Superiority; Regression, Linear; Analysis performed using linear regression ANCOVA with covariates of Baseline potassium, gender, age and treatment; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.26 to 0.34]

26. Secondary Outcome: Mean Weighted Mean 0-4 h of Glucose and Potassium, Maximum Glucose 0-4 h and Minimum Potassium 0-4 h Over Time
Description: Blood samples were collected at pre-dose and 4 h post-dose on Day 1, Day 2, Day 7, Day 8, Day 14 and Day 15. Weighted mean was calculated by calculating the AUC, and then dividing by the relevant time interval. AUC was calculated using the trapezoidal rule.
Time Frame: Day 1 up to Day 15
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17 | 16 | 17 | 18
mmol/L
  Weighted Mean Glucose 0-4 h, Day 1: number analyzed (Participants) | 16 | 16 | 16 | 17
  Weighted Mean Glucose 0-4 h, Day 1 | 5.917 (1.4350) | 5.202 (0.6244) | 5.537 (0.8241) | 5.744 (1.0359)
  Weighted Mean Glucose 0-4 h, Day 2: number analyzed (Participants) | 15 | 15 | 15 | 16
  Weighted Mean Glucose 0-4 h, Day 2 | 5.913 (1.4064) | 5.237 (1.0555) | 5.763 (1.1516) | 5.626 (1.3748)
  Weighted Mean Glucose 0-4 h, Day 7: number analyzed (Participants) | 16 | 15 | 11 | 15
  Weighted Mean Glucose 0-4 h, Day 7 | 5.860 (1.0459) | 5.271 (0.6604) | 5.636 (1.0571) | 5.649 (1.2134)
  Weighted Mean Glucose 0-4 h, Day 8: number analyzed (Participants) | 16 | 14 | 11 | 14
  Weighted Mean Glucose 0-4 h, Day 8 | 5.679 (1.4463) | 5.266 (0.9408) | 5.839 (1.5742) | 5.461 (1.2427)
  Weighted Mean Glucose 0-4 h, Day 14: number analyzed (Participants) | 15 | 14 | 11 | 14
  Weighted Mean Glucose 0-4 h, Day 14 | 6.035 (1.1987) | 5.406 (0.4841) | 5.384 (0.6367) | 5.460 (0.8837)
  Weighted Mean Glucose 0-4 h, Day 15: number analyzed (Participants) | 15 | 15 | 12 | 14
  Weighted Mean Glucose 0-4 h, Day 15 | 5.927 (1.3819) | 5.196 (0.8684) | 5.599 (1.1422) | 5.557 (1.2105)
  Weighted Mean Potassium 0-4 h, Day 1: number analyzed (Participants) | 16 | 13 | 15 | 13
  Weighted Mean Potassium 0-4 h, Day 1 | 4.491 (0.5698) | 4.271 (0.6109) | 4.174 (0.3005) | 4.352 (0.3550)
  Weighted Mean Potassium 0-4 h, Day 2: number analyzed (Participants) | 14 | 14 | 14 | 14
  Weighted Mean Potassium 0-4 h, Day 2 | 4.645 (0.5498) | 4.541 (0.3952) | 4.220 (0.2719) | 4.628 (0.8501)
  Weighted Mean Potassium 0-4 h, Day 7: number analyzed (Participants) | 15 | 13 | 10 | 13
  Weighted Mean Potassium 0-4 h, Day 7 | 4.494 (0.8933) | 4.212 (0.4412) | 4.154 (0.3908) | 4.258 (0.4597)
  Weighted Mean Potassium 0-4 h, Day 8: number analyzed (Participants) | 15 | 14 | 10 | 12
  Weighted Mean Potassium 0-4 h, Day 8 | 4.525 (0.4862) | 4.549 (0.4950) | 4.240 (0.3727) | 4.503 (0.3247)
  Weighted Mean Potassium 0-4 h, Day 14: number analyzed (Participants) | 15 | 13 | 11 | 12
  Weighted Mean Potassium 0-4 h, Day 14 | 4.458 (0.5101) | 4.298 (0.5123) | 4.250 (0.3694) | 4.321 (0.2958)
  Weighted Mean Potassium 0-4 h, Day 15: number analyzed (Participants) | 15 | 14 | 12 | 12
  Weighted Mean Potassium 0-4 h, Day 15 | 4.400 (0.4552) | 4.582 (0.3869) | 4.241 (0.4811) | 4.466 (0.2841)
  Maximum Glucose 0-4 h, Day 1 | 6.62 (2.434) | 5.54 (0.801) | 6.11 (1.582) | 6.12 (1.235)
  Maximum Glucose 0-4 h, Day 2: number analyzed (Participants) | 16 | 16 | 17 | 17
  Maximum Glucose 0-4 h, Day 2 | 6.29 (1.735) | 5.77 (1.411) | 6.21 (1.439) | 6.13 (1.728)
  Maximum Glucose 0-4 h, Day 7: number analyzed (Participants) | 16 | 15 | 13 | 15
  Maximum Glucose 0-4 h, Day 7 | 6.49 (1.539) | 5.60 (0.967) | 6.24 (2.103) | 6.28 (1.560)
  Maximum Glucose 0-4 h, Day 8: number analyzed (Participants) | 16 | 15 | 13 | 14
  Maximum Glucose 0-4 h, Day 8 | 6.16 (1.990) | 5.64 (0.993) | 6.25 (1.850) | 6.14 (1.914)
  Maximum Glucose 0-4 h, Day 14: number analyzed (Participants) | 16 | 15 | 13 | 14
  Maximum Glucose 0-4 h, Day 14 | 6.30 (1.477) | 5.67 (0.976) | 6.50 (2.724) | 5.86 (1.241)
  Maximum Glucose 0-4 h, Day 15: number analyzed (Participants) | 16 | 15 | 12 | 14
  Maximum Glucose 0-4 h, Day 15 | 6.28 (1.636) | 5.61 (1.113) | 6.37 (1.592) | 6.19 (1.664)
  Minimum Potassium 0-4 h, Day 1: number analyzed (Participants) | 17 | 15 | 17 | 16
  Minimum Potassium 0-4 h, Day 1 | 4.18 (0.427) | 4.05 (0.584) | 4.02 (0.307) | 3.94 (0.341)
  Minimum Potassium 0-4 h, Day 2: number analyzed (Participants) | 16 | 15 | 17 | 15
  Minimum Potassium 0-4 h, Day 2 | 4.35 (0.346) | 4.24 (0.412) | 4.03 (0.291) | 4.28 (0.810)
  Minimum Potassium 0-4 h, Day 7: number analyzed (Participants) | 16 | 14 | 13 | 13
  Minimum Potassium 0-4 h, Day 7 | 4.28 (0.835) | 3.91 (0.501) | 3.89 (0.355) | 3.91 (0.535)
  Minimum Potassium 0-4 h, Day 8: number analyzed (Participants) | 16 | 14 | 13 | 12
  Minimum Potassium 0-4 h, Day 8 | 4.34 (0.468) | 4.34 (0.473) | 4.00 (0.338) | 4.28 (0.328)
  Minimum Potassium 0-4 h, Day 14: number analyzed (Participants) | 16 | 14 | 13 | 12
  Minimum Potassium 0-4 h, Day 14 | 4.20 (0.388) | 4.15 (0.467) | 4.00 (0.163) | 4.08 (0.376)
  Minimum Potassium 0-4 h, Day 15: number analyzed (Participants) | 16 | 14 | 12 | 12
  Minimum Potassium 0-4 h, Day 15 | 4.24 (0.430) | 4.29 (0.366) | 3.93 (0.379) | 4.22 (0.279)

27. Secondary Outcome: AUC of GW642444H Over 0 to 4 h (AUC [0-4]) on Day 1, 7 and 14
Description: Blood samples were collected on Day 1 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose), Day 7 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose) and Day 14 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose). The pre-dose sample was collected within 5 min prior to study medication administration. The AUC over 4 h as AUC from zero (pre-dose) to 2 h post-dose (AUC [0-2]), AUC from zero (pre-dose) to 4 h post-dose (AUC [0-4]) and AUC from zero (pre-dose) to time of last quantifiable concentration (AUC [0-t]) was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: Day 1 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose), Day 7 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose) and Day 14 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose)
Population: Pharmacokinetic (PK) Concentration Population comprised of those participants in the Safety Population for whom a PK sample was obtained and analyzed. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram (pg)*h/mL
Arm/Group | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily
Number analyzed (Participants) | 16 | 16
Picogram (pg)*h/mL
  AUC (0-2), Day 1: number analyzed (Participants) | 6 | 16
  AUC (0-2), Day 1 | 151.067 (39.92) | NA (NA) — AUC0-2 was not calculated for GW642444 400 mcg once daily.
  AUC (0-2), Day 7: number analyzed (Participants) | 8 | 16
  AUC (0-2), Day 7 | 164.374 (57.30) | NA (NA) — AUC0-2 was not calculated for GW642444 400 mcg once daily.
  AUC (0-2), Day 14: number analyzed (Participants) | 10 | 16
  AUC (0-2), Day 14 | 166.055 (40.98) | NA (NA) — AUC0-2 was not calculated for GW642444 400 mcg once daily.
  AUC (0-4), Day 1: number analyzed (Participants) | 4 | 14
  AUC (0-4), Day 1 | 277.582 (14.92) | 699.719 (60.50)
  AUC (0-4), Day 7: number analyzed (Participants) | 4 | 11
  AUC (0-4), Day 7 | 412.496 (31.95) | 945.893 (58.35)
  AUC (0-4), Day 14: number analyzed (Participants) | 9 | 11
  AUC (0-4), Day 14 | 300.921 (40.05) | 772.694 (35.59)
  AUC (0-t), Day 1: number analyzed (Participants) | 8 | 14
  AUC (0-t), Day 1 | 192.799 (51.42) | 702.937 (60.22)
  AUC (0-t), Day 7: number analyzed (Participants) | 8 | 13
  AUC (0-t), Day 7 | 212.547 (86.45) | 840.634 (63.50)
  AUC (0-t), Day 14: number analyzed (Participants) | 10 | 12
  AUC (0-t), Day 14 | 275.621 (49.02) | 736.842 (40.06)

28. Secondary Outcome: Maximum Concentration (Cmax) of GW642444H at Day 1, 7 and 14
Description: Blood samples were collected on Day 1 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose), Day 7 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose) and Day 14 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose). The pre-dose sample was collected within 5 min prior to study medication administration. The first occurrence of the Cmax was determined directly from the raw concentration-time data.
Time Frame: as for outcome 27
Population: PK Concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily
Number analyzed (Participants) | 16 | 16
pg/mL
  Day 1 | 78.851 (45.85) | 226.407 (108.53)
  Day 7: number analyzed (Participants) | 14 | 13
  Day 7 | 82.642 (64.09) | 427.282 (49.41)
  Day 14: number analyzed (Participants) | 14 | 12
  Day 14 | 92.089 (50.15) | 308.546 (24.25)

29. Secondary Outcome: Time to Maximum Concentration (Tmax) and Time of Last Quantifiable Concentration (Tlast) of GW642444H at Day 1, 7 and 14
Description: Blood samples were collected on Day 1 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose), Day 7 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose) and Day 14 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose). The pre-dose sample was collected within 5 min prior to study medication administration. The time at which Cmax was observed and tlast was determined directly from the raw concentration-time data.
Time Frame: as for outcome 27
Population: PK Concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: h
Arm/Group | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily
Number analyzed (Participants) | 16 | 16
h
  Tmax, Day 1 | 1.000 [0.08 to 4.00] | 1.000 [0.08 to 1.08]
  Tmax, Day 7: number analyzed (Participants) | 14 | 13
  Tmax, Day 7 | 1.000 [0.08 to 4.00] | 0.130 [0.08 to 1.02]
  Tmax, Day 14: number analyzed (Participants) | 14 | 12
  Tmax, Day 14 | 0.555 [0.08 to 2.00] | 0.525 [0.07 to 2.02]
  Tlast, Day 1 | 2.000 [0.98 to 4.00] | 4.000 [0.08 to 4.23]
  Tlast, Day 7: number analyzed (Participants) | 13 | 13
  Tlast, Day 7 | 2.000 [1.00 to 4.00] | 4.000 [1.97 to 4.17]
  Tlast, Day 14: number analyzed (Participants) | 14 | 12
  Tlast, Day 14 | 4.000 [0.08 to 4.12] | 4.000 [2.00 to 4.88]

30. Secondary Outcome: AUC (0-4) of CCI2189 at Day 1, 7 and 14
Description: CCI2189 is a counterion of GW642444H. Blood samples were collected on Day 1 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose), Day 7 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose) and Day 14 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose). The pre-dose sample was collected within 5 min prior to study medication administration. The AUC (0-4) was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: as for outcome 27
Population: PK Concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram (ng)*h/mL
Arm/Group | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily
Number analyzed (Participants) | 16 | 16
Nanogram (ng)*h/mL
  Day 1: number analyzed (Participants) | 16 | 14
  Day 1 | 11.779 (34.10) | 45.664 (25.35)
  Day 7: number analyzed (Participants) | 12 | 12
  Day 7 | 12.155 (33.83) | 52.866 (41.09)
  Day 14: number analyzed (Participants) | 13 | 11
  Day 14 | 13.683 (34.35) | 48.348 (36.69)

31. Secondary Outcome: Cmax of CCI2189 at Day 1, 7 and 14
Description: CCI2189 is a counterion of GW642444H. Blood samples were collected on Day 1 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose), Day 7 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose) and Day 14 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose). The pre-dose sample was collected within 5 min prior to study medication administration. The first occurrence of the Cmax was determined directly from the raw concentration-time data.
Time Frame: as for outcome 27
Population: PK Concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily
Number analyzed (Participants) | 16 | 16
ng/mL
  Day 1: number analyzed (Participants) | 16 | 15
  Day 1 | 4.692 (34.06) | 15.650 (55.22)
  Day 7: number analyzed (Participants) | 14 | 13
  Day 7 | 4.578 (27.23) | 21.293 (37.74)
  Day 14: number analyzed (Participants) | 14 | 12
  Day 14 | 5.115 (34.66) | 18.315 (28.69)

32. Secondary Outcome: AUC (0-4) of GW630200 and GSK932009 at Day 1, 7 and 14
Description: GW630200 and GSK932009 are metabolites of GW642444H. Blood samples were collected on Day 1 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose), Day 7 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose) and Day 14 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose). The pre-dose sample was collected within 5 min prior to study medication administration. The AUC (0-4) was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: as for outcome 27
Population: PK Concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily
Number analyzed (Participants) | 16 | 16
pg*h/mL
  GW630200, Day 1 | NA (NA) — Data was not quantifiable. | NA (NA) — Data was not quantifiable.
  GW630200, Day 7 | NA (NA) — Data was not quantifiable. | NA (NA) — Data was not quantifiable.
  GW630200, Day 14 | NA (NA) — Data was not quantifiable. | NA (NA) — Data was not quantifiable.
  GSK932009, Day 1: number analyzed (Participants) | 0 | 5
  GSK932009, Day 1 |  | 1222.771 (19.18)
  GSK932009, Day 7: number analyzed (Participants) | 1 | 7
  GSK932009, Day 7 | 897.695 (NA) — Only one participant was analyzed. | 1866.738 (58.04)
  GSK932009, Day 14: number analyzed (Participants) | 1 | 5
  GSK932009, Day 14 | 797.075 (NA) — Only one participant was analyzed. | 1527.671 (20.22)

33. Secondary Outcome: Cmax of GW630200 and GSK932009 at Day 1, 7 and 14
Description: GW630200 and GSK932009 are metabolites of GW642444H. Blood samples were collected on Day 1 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose), Day 7 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose) and Day 14 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose). The pre-dose sample was collected within 5 min prior to study medication administration. The first occurrence of the Cmax was determined directly from the raw concentration-time data.
Time Frame: as for outcome 27
Population: PK Concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily
Number analyzed (Participants) | 16 | 16
pg/mL
  GW630200, Day 1 | NA (NA) — Data was not quantifiable. | NA (NA) — Data was not quantifiable.
  GW630200, Day 7 | NA (NA) — Data was not quantifiable. | NA (NA) — Data was not quantifiable.
  GW630200, Day 14 | NA (NA) — Data was not quantifiable. | NA (NA) — Data was not quantifiable.
  GSK932009, Day 1: number analyzed (Participants) | 0 | 13
  GSK932009, Day 1 |  | 311.740 (36.96)
  GSK932009, Day 7: number analyzed (Participants) | 2 | 12
  GSK932009, Day 7 | 235.459 (17.81) | 460.352 (69.16)
  GSK932009, Day 14: number analyzed (Participants) | 2 | 12
  GSK932009, Day 14 | 228.419 (19.25) | 391.680 (37.49)

34. Secondary Outcome: Time to Maximum Concentration (Tmax) of CCI2189, GW630200 and GSK932009 at Day 1, 7 and 14
Description: GW630200 and GSK932009 are metabolites of GW642444H. CCI2189 is a counterion of GW642444H. Blood samples were collected on Day 1 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose), Day 7 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose) and Day 14 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose). The pre-dose sample was collected within 5 min prior to study medication administration. The time at which Cmax was observed was determined directly from the raw concentration-time data.
Time Frame: as for outcome 27
Population: PK Concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: h
Arm/Group | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily
Number analyzed (Participants) | 16 | 16
h
  CC12189, Day 1: number analyzed (Participants) | 16 | 15
  CC12189, Day 1 | 1.285 [0.93 to 4.00] | 1.000 [0.08 to 4.00]
  CC12189, Day 7: number analyzed (Participants) | 14 | 13
  CC12189, Day 7 | 1.010 [0.95 to 4.00] | 1.000 [0.10 to 2.00]
  CC12189, Day 14: number analyzed (Participants) | 14 | 12
  CC12189, Day 14 | 1.000 [0.08 to 4.00] | 1.000 [0.07 to 4.00]
  GW630200, Day 1 | NA [NA to NA] — Data was not quantifiable. | NA [NA to NA] — Data was not quantifiable.
  GW630200, Day 7 | NA [NA to NA] — Data was not quantifiable. | NA [NA to NA] — Data was not quantifiable.
  GW630200, Day 14 | NA [NA to NA] — Data was not quantifiable. | NA [NA to NA] — Data was not quantifiable.
  GSK932009, Day 1: number analyzed (Participants) | 0 | 16
  GSK932009, Day 1 |  | 2.050 [1.00 to 4.23]
  GSK932009, Day 7: number analyzed (Participants) | 2 | 12
  GSK932009, Day 7 | 2.500 [1.00 to 4.00] | 2.000 [1.00 to 4.00]
  GSK932009, Day 14: number analyzed (Participants) | 2 | 12
  GSK932009, Day 14 | 1.500 [1.00 to 2.00] | 2.000 [1.00 to 4.00]

35. Secondary Outcome: AUC (0-4) of Salmeterol at Day 1, 7 and 14
Description: Blood samples were collected on Day 1 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose), Day 7 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose) and Day 14 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose). The pre-dose sample was collected within 5 min prior to study medication administration. The AUC (0-4) was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: as for outcome 27
Population: PK Concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17
pg*h/mL
  Day 1: number analyzed (Participants) | 4
  Day 1 | 225.334 (14.83)
  Day 7: number analyzed (Participants) | 8
  Day 7 | 226.708 (34.42)
  Day 14: number analyzed (Participants) | 6
  Day 14 | 178.656 (33.47)

36. Secondary Outcome: Cmax of Salmeterol at Day 1, 7 and 14
Description: as for outcome 28
Time Frame: as for outcome 27
Population: PK Concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17
pg*h/mL
  Day 1: number analyzed (Participants) | 15
  Day 1 | 50.218 (45.71)
  Day 7: number analyzed (Participants) | 12
  Day 7 | 59.943 (49.73)
  Day 14: number analyzed (Participants) | 11
  Day 14 | 51.983 (29.13)

37. Secondary Outcome: Tmax of Salmeterol at Day 1, 7 and 14
Description: Blood samples were collected on Day 1 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose), Day 7 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose) and Day 14 (pre-dose, 5 min, 1 h, 2 h and 4 h post-dose). The pre-dose sample was collected within 5 min prior to study medication administration. The time at which Cmax was observed was determined directly from the raw concentration-time data.
Time Frame: as for outcome 27
Population: PK Concentration Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: h
Arm/Group | Salmeterol 50 mcg BD
Number analyzed (Participants) | 17
h
  Day 1: number analyzed (Participants) | 15
  Day 1 | 1.000 [0.08 to 2.00]
  Day 7: number analyzed (Participants) | 12
  Day 7 | 1.000 [0.08 to 2.00]
  Day 14: number analyzed (Participants) | 11
  Day 14 | 1.000 [0.08 to 4.05]

ADVERSE EVENTS:
Time Frame: AEs were collected up to Follow-up (17 days)
Description: Safety Population was used.
Arm/Group | Placebo | GW642444 100 mcg Once Daily | GW642444 400 mcg Once Daily | Salmeterol 50 mcg BD
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 1/17 | 1/18
Other Adverse Events (participants affected / at risk) | 4/17 | 5/16 | 7/17 | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | GW642444 100 mcg Once Daily (N=16) | GW642444 400 mcg Once Daily (N=17) | Salmeterol 50 mcg BD (N=18)
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | GW642444 100 mcg Once Daily (N=16) | GW642444 400 mcg Once Daily (N=17) | Salmeterol 50 mcg BD (N=18)
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 2 | 2 | 4 | 3
Tension headache (Nervous system disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 2 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 1
Application site rash (General disorders) | 1 | 0 | 0 | 0
Application site reaction (General disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.